CLINICAL TRIAL: NCT04982445
Title: A Phase 4, Open-label, Single Arm Study to Optimize Implementation of CABENUVA for the Treatment of HIV-1, for Administration in U.S. Community-based Infusion Centers or Other Alternate Sites of Administration
Brief Title: Study Using CABENUVA™ for the Treatment of Human Immunodeficiency Virus (HIV)-1, Administered in Infusion Centers (IC) or Alternate Sites of Administration (ASA) in the United States (U.S.)
Acronym: GLACIER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 214747
Record Dates: First submitted 2021-07-26; First posted 2021-07-29 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: HIV Infections
Keywords: HIV; CABENUVA; Intramuscular; Cabotegravir; Rilpivirine
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir, rilpivirine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants receiving CABENUVA (Experimental): Eligible participants received CABENUVA injections intramuscularly at infusion centers/ASAs monthly or every-2-months.
  Interventions: Drug: CABENUVA

INTERVENTIONS:
Drug: CABENUVA — CABENUVA will be administered IM at infusion centers/ASAs

SUMMARY:
GLACIER (Giving Long Acting CABENUVA in an Infusion center/ASA) is an interventional study examining the administration of CABENUVA (Cabotegravir long acting [LA] plus Rilpivirine LA) intramuscular (IM) in infusion centers/ASAs in United States. In this study, the intervention is the process of using an infusion center/ASA as the location to receive the CABENUVA IM injections. The acceptability and feasibility of the IC/ASA to deliver CABENUVA IM injections will be assessed from the perspectives of the participants, HIV care providers and IC/ASA staff. In this study, Month 1 is the Baseline visit. CABENUVA is a registered trademark of ViiV Healthcare.

ELIGIBILITY:
Inclusion criteria

* Adults (greater than or equal to [>=]18 years old) at the time of signing the informed consent.
* HIV-1 infected and have been prescribed CABNEUVA per the United States Prescribing information (USPI).
* Participants can be enrolled
* If they have been taking oral VOCABRIA + EDURANT or other ART for approximately 1 month (at least 28 days) prior to Baseline/Month 1, or
* Already taking CABENUVA prior to Baseline/Month 1 and the last injections were within a 1 month +/- 7-day window or for every 2-month injections, the timing will vary if they are receiving the initiation injections (1 month +/- 7-day) or the continuation injections (2 months +/- 7 days) per the USPI, or
* Prescribed direct to inject and receive their 1st injection without an oral lead in at the Infusion Center/ASA on the last day of any other antiretroviral therapy
* Agreement to receive CABENUVA IM injections at participating infusion center/ASA.

Exclusion criteria

* Participants are excluded from the study as dictated in the Prescribing Information (CABENUVA [USPI]) in consultation with the HIV care provider.
* Contraindications, as per the current Prescribing Information [CABENUVA USPI]
* New health condition / prohibited medication reported - Other Reason at the discretion of the HIV care provider or IC/ ASA staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (15):
- United States (15):
  - GSK Investigational Site, Evans, Georgia
  - GSK Investigational Site, East Lansing, Michigan
  - GSK Investigational Site, Novi, Michigan
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Florence, South Carolina
  - GSK Investigational Site, Summerville, South Carolina
  - GSK Investigational Site, West Columbia, South Carolina
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Kingwood, Texas
  - GSK Investigational Site, North Richland Hills, Texas
  - GSK Investigational Site, Plano, Texas

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 44 patients living with HIV (PLWHIV) were enrolled in the study and all of them received study treatment and were included in the safety population. Staff such as HIV care providers and IC/ ASA staff were not counted as enrolled.
Period: Overall Study
Arm/Group | Participants Receiving CABENUVA
Started | 44
Completed | 38
Not Completed | 6
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.8 (12.64)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 35
  Female | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Agree or Completely Agree (a Score of 4 or Higher) Across All Items on the Feasibility of Intervention Measure (FIM)
Description: Feasibility of Intervention Measure (FIM) were employed to evaluate the feasibility of CABENUVA administration at Infusion Centers (IC)/ alternate sites of administration (ASA). Higher scores on FIM indicate greater feasibility, where each item can be scored from 1 to 5: Completely disagree (score=1), disagree (score=2), neither agree or disagree (score=3), agree (score=4), completely agree (score=5). This scoring looked at the number responding '4' or '5' to each question divided by the number completing all 4-items where "items" refer to the individual questions or statements that participants respond to in order to assess their perceptions of an intervention. Each item is designed to measure a specific aspect of either acceptability or feasibility.
Time Frame: At Month 8
Population: Analysis was performed on the Safety set which includes any participant who completed any portion of any questionnaire at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 37
Participants | 31

2. Secondary Outcome: Number of Participants Who Agree or Completely Agree (a Score of 4 or Higher) Across All Items on the FIM at Month 1 and 3
Time Frame: At Months 1 and 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 43
Participants
  Month 1 | 37
  Month 3: number analyzed (Participants) | 36
  Month 3 | 31

3. Secondary Outcome: Number of HIV Care Providers Who Agree or Completely Agree (a Score of 4 or Higher) Across All Items on the FIM at Month 1, 4 and 8
Time Frame: At Months 1, 4, and 8
Population: Analysis was performed on the HIV care providers which includes any HIV care provider who completed any portion of any questionnaire at the specified timepoint.
Measure: Count of Participants; unit: Participants
Groups:
- HIV Care Providers: Eligible HIV Care Providers completed study assessments at each data collection time point.
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 3
Participants
  Month 1 | 1
  Month 4 | 1
  Month 8: number analyzed (Participants) | 2
  Month 8 | 0

4. Secondary Outcome: Number of IC/ ASA Staff Who Agree or Completely Agree (a Score of 4 or Higher) Across All Items on the FIM Prior to Month 1 and at Months 3 and 8
Time Frame: Prior to Month 1 (Baseline) and at Months 3 and 8
Population: Analysis was performed on the IC/ASA staff which includes any IC/ASA staff who completed any portion of any questionnaire at the specified timepoint.
Measure: Count of Participants; unit: Participants
Groups:
- IC/ASA Staff: Eligible IC/ASA Staff completed study assessments at each data collection time point.
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 113
Participants
  Prior to Month 1 (Baseline) | 50
  Month 3: number analyzed (Participants) | 34
  Month 3 | 19
  Month 8: number analyzed (Participants) | 19
  Month 8 | 11

5. Secondary Outcome: Change in FIM Score Over Time in Participants at Month 3 and 8
Description: The mean score for feasibility of the intervention administration was calculated by averaging the responses from the 4 items. The responses were scored based on a scale of 1 to 5 where 1=completely disagree, 2=disagree, 3=neither agree nor disagree, 4=agree, and 5=completely agree.
Time Frame: From Month 1 (Baseline) to Months 3 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 36
Scores on a scale
  From Baseline to Month 3: number analyzed (Participants) | 35
  From Baseline to Month 3 | 0.06 (0.667)
  From Baseline to Month 8 | -0.03 (0.677)

6. Secondary Outcome: Change in FIM Score Over Time in HIV Care Providers at Month 4 and 8
Time Frame: From Month 1 (Baseline) to Months 4 and 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 3
Scores on a scale
  From Baseline to Month 4 | 0.33 (0.764)
  From Baseline to Month 8: number analyzed (Participants) | 2
  From Baseline to Month 8 | 0.38 (0.177)

7. Secondary Outcome: Change in FIM Score Over Time in IC/ ASA Staff at Month 3 and 8
Time Frame: From Month 1 (Baseline) to Months 3 and 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 34
Scores on a scale
  From Baseline to Month 3 | -0.04 (0.729)
  From Baseline to Month 8: number analyzed (Participants) | 20
  From Baseline to Month 8 | -0.20 (0.700)

8. Secondary Outcome: Number of Participants Assessed for Feasibility of CABENUVA Administration by Other Quantitative Questionnaires at Month 1
Description: The tailored questionnaire for participants receiving CABENUVA was developed specifically for this study and contains items regarding the reasons for switching to CABENUVA, adherence to their previous oral HIV medication, preferences and attitudes regarding their medication regimen, and perceived advantages and disadvantages of receiving injections at the IC/ASA. In this outcome measure, participants were asked about their views on the IC/ASA administration model (any/biggest concerns about receiving CABENUVA at an infusion center).
Time Frame: At Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 44
Participants
  No current worries about receiving CABENUVA at an infusion center | 19
  Scheduling upcoming CABENUVA visits | 7
  Forgetting my appointments for the CABENUVA visits | 6
  My doctor not knowing if I have a bad reaction | 4
  Other | 4
  The infusion center managing my pain or soreness from CABENUVA | 3
  The infusion center managing the side effects from CABENUVA | 3
  The infusion center not aware of my other medical history | 3
  Transportation to the infusion center for the CABENUVA visits | 3
  The infusion center hours for CABENUVA visits | 3
  Others at the clinic may find out that I am HIV positive | 3
  Frequency of the required visits to the infusion center clinic as well as my primary HIV doctor | 2
  Rescheduling missed CABENUVA visits | 1
  Infusion center not aware of my other medications and possible interactions | 0
  Parking at the infusion center for CABENUVA visits | 0
  Childcare during CABENUVA visits | 0
  Infusion center not being an HIV-specific clinic | 0
  Missing | 1

9. Secondary Outcome: Number of Participants Assessed for Feasibility of CABENUVA Administration (Concern About Continuing to Receive CABENUVA) by Other Quantitative Questionnaires at Month 3 and 8
Description: The tailored questionnaire for participants receiving CABENUVA was developed specifically for this study and contains items regarding the reasons for switching to CABENUVA, adherence to their previous oral HIV medication, preferences and attitudes regarding their medication regimen, and perceived advantages and disadvantages of receiving injections at the IC/ASA. In this outcome measure, participants were asked about their views on the IC/ASA administration model (any concerns about continuing to receive CABENUVA at an infusion center) at Months 3 and 8.
Time Frame: At Month 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 41
Participants
  Month 3- Do you have any concerns about continuing to receive CABENUVA at an infusion center?: Yes | 3
  Month 3- Do you have any concerns about continuing to receive CABENUVA at an infusion center?: No | 33
  Month 3- Do you have any concerns about continuing to receive CABENUVA at an infusion center?: Missing | 5
  Month 8- Do you have any concerns about continuing to receive CABENUVA at an infusion center?: number analyzed (Participants) | 38
  Month 8- Do you have any concerns about continuing to receive CABENUVA at an infusion center?: Yes | 3
  Month 8- Do you have any concerns about continuing to receive CABENUVA at an infusion center?: No | 34
  Month 8- Do you have any concerns about continuing to receive CABENUVA at an infusion center?: Missing | 1

10. Secondary Outcome: Number of Participants Assessed for Feasibility of CABENUVA Administration by Other Quantitative Questionnaires at Month 3 and 8
Description: Participants were asked about their views on the IC/ASA administration model (biggest concerns about continuing to receive CABENUVA at an infusion center).
Time Frame: At Month 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 41
Participants
  Month 3- The infusion center managing my pain or soreness from CABENUVA | 1
  Month 3- The infusion center managing the side effects from CABENUVA: number analyzed (Participants) | 3
  Month 3- The infusion center managing the side effects from CABENUVA | 1
  Month 3- My doctor not knowing if I have a bad reaction | 1
  Month 3- Scheduling upcoming CABENUVA visits | 1
  Month 3- Transportation to the infusion center for the CABENUVA visits | 1
  Month 3- Others at the clinic may find out that I am HIV positive | 1
  Month 3- Other | 1
  Month 3- The infusion center not aware of my other medical history | 0
  Month 3- Infusion center not aware of my other medications and possible interactions | 0
  Month 3- Rescheduling missed CABENUVA visits | 0
  Month 3- Forgetting my appointments for the CABENUVA visits | 0
  Month 3- Frequency of the required visits to infusion center clinic as well as my primary HIV doctor | 0
  Month 3- Parking at the infusion center for CABENUVA visits | 0
  Month 3- The infusion center hours for CABENUVA visits | 0
  Month 3- Childcare during CABENUVA visits | 0
  Month 3- Infusion center not being an HIV-specific clinic | 0
  Month 3- Missing | 5
  Month 8- The infusion center managing my pain or soreness from CABENUVA: number analyzed (Participants) | 38
  Month 8- The infusion center managing my pain or soreness from CABENUVA | 0
  Month 8- The infusion center managing the side effects from CABENUVA: number analyzed (Participants) | 38
  Month 8- The infusion center managing the side effects from CABENUVA | 0
  Month 8- My doctor not knowing if I have a bad reaction: number analyzed (Participants) | 38
  Month 8- My doctor not knowing if I have a bad reaction | 0
  Month 8- Scheduling upcoming CABENUVA visits: number analyzed (Participants) | 38
  Month 8- Scheduling upcoming CABENUVA visits | 0
  Month 8- Transportation to the infusion center for the CABENUVA visits: number analyzed (Participants) | 38
  Month 8- Transportation to the infusion center for the CABENUVA visits | 0
  Month 8- Others at the clinic may find out that I am HIV positive: number analyzed (Participants) | 38
  Month 8- Others at the clinic may find out that I am HIV positive | 0
  Month 8- Other: number analyzed (Participants) | 38
  Month 8- Other | 3
  Month 8- The infusion center not aware of my other medical history: number analyzed (Participants) | 38
  Month 8- The infusion center not aware of my other medical history | 0
  Month 8- Infusion center not aware of my other medications and possible interactions: number analyzed (Participants) | 38
  Month 8- Infusion center not aware of my other medications and possible interactions | 0
  Month 8- Rescheduling missed CABENUVA visits: number analyzed (Participants) | 38
  Month 8- Rescheduling missed CABENUVA visits | 0
  Month 8- Forgetting my appointments for the CABENUVA visits: number analyzed (Participants) | 38
  Month 8- Forgetting my appointments for the CABENUVA visits | 0
  Month 8- Frequency of the required visits to infusion center clinic as well as my primary HIV doctor: number analyzed (Participants) | 38
  Month 8- Frequency of the required visits to infusion center clinic as well as my primary HIV doctor | 0
  Month 8- Parking at the infusion center for CABENUVA visits: number analyzed (Participants) | 38
  Month 8- Parking at the infusion center for CABENUVA visits | 0
  Month 8- The infusion center hours for CABENUVA visits: number analyzed (Participants) | 38
  Month 8- The infusion center hours for CABENUVA visits | 0
  Month 8- Childcare during CABENUVA visits: number analyzed (Participants) | 38
  Month 8- Childcare during CABENUVA visits | 0
  Month 8- Infusion center not being an HIV-specific clinic: number analyzed (Participants) | 38
  Month 8- Infusion center not being an HIV-specific clinic | 0
  Month 8- Missing: number analyzed (Participants) | 38
  Month 8- Missing | 1

11. Secondary Outcome: Number of HIV Care Providers Assessed for Feasibility of CABENUVA Administration in Participants by Other Quantitative Questionnaires at Month 1
Description: The tailored HIV care provider/clinical staff questionnaire was developed specifically for this study and contains items regarding the provider's practice and experience, as well as their attitudes, expectations, and concerns regarding the use of CABENUVA/long-acting injectable administered by ICs/ASAs.
Time Frame: At Month 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 3
Participants
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Extremely concerned | 1
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Moderately concerned | 1
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Somewhat concerned | 1
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Slightly concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Not at all concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Missing | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Extremely concerned | 1
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Moderately concerned | 1
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Somewhat concerned | 1
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Slightly concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Not at all concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Missing | 0
  Patients not being virologically suppressed due to missed injections: Extremely concerned | 0
  Patients not being virologically suppressed due to missed injections: Moderately concerned | 2
  Patients not being virologically suppressed due to missed injections: Somewhat concerned | 1
  Patients not being virologically suppressed due to missed injections: Slightly concerned | 0
  Patients not being virologically suppressed due to missed injections: Not at all concerned | 0
  Patients not being virologically suppressed due to missed injections: Missing | 0
  Being informed (in a timely manner) of adverse events: Extremely concerned | 0
  Being informed (in a timely manner) of adverse events: Moderately concerned | 2
  Being informed (in a timely manner) of adverse events: Somewhat concerned | 1
  Being informed (in a timely manner) of adverse events: Slightly concerned | 0
  Being informed (in a timely manner) of adverse events: Not at all concerned | 0
  Being informed (in a timely manner) of adverse events: Missing | 0
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Extremely concerned | 0
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Moderately concerned | 2
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Somewhat concerned | 0
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Slightly concerned | 1
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Not at all concerned | 0
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Missing | 0

12. Secondary Outcome: Number of HIV Care Providers Assessed for Feasibility of CABENUVA Administration in Participants by Other Quantitative Questionnaires at Month 4
Time Frame: At Month 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 3
Participants
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Extremely concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Moderately concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Somewhat concerned | 3
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Slightly concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Not at all concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Missing | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Extremely concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Moderately concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Somewhat concerned | 3
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Slightly concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Not at all concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Missing | 0
  Patients not being virologically suppressed due to missed injections: Extremely concerned | 0
  Patients not being virologically suppressed due to missed injections: Moderately concerned | 2
  Patients not being virologically suppressed due to missed injections: Somewhat concerned | 0
  Patients not being virologically suppressed due to missed injections: Slightly concerned | 1
  Patients not being virologically suppressed due to missed injections: Not at all concerned | 0
  Patients not being virologically suppressed due to missed injections: Missing | 0
  Being informed (in a timely manner) of adverse events: Extremely concerned | 0
  Being informed (in a timely manner) of adverse events: Moderately concerned | 1
  Being informed (in a timely manner) of adverse events: Somewhat concerned | 1
  Being informed (in a timely manner) of adverse events: Slightly concerned | 1
  Being informed (in a timely manner) of adverse events: Not at all concerned | 0
  Being informed (in a timely manner) of adverse events: Missing | 0
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Extremely concerned | 1
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Moderately concerned | 0
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Somewhat concerned | 1
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Slightly concerned | 1
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Not at all concerned | 0
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Missing | 0

13. Secondary Outcome: Number of HIV Care Providers Assessed for Feasibility of CABENUVA Administration in Participants by Other Quantitative Questionnaires at Month 8
Time Frame: At Month 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 3
Participants
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Extremely concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Moderately concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Somewhat concerned | 1
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Slightly concerned | 1
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Not at all concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Missing | 1
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Extremely concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Moderately concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Somewhat concerned | 1
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Slightly concerned | 1
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Not at all concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Missing | 1
  Patients not being virologically suppressed due to missed injections: Extremely concerned | 0
  Patients not being virologically suppressed due to missed injections: Moderately concerned | 0
  Patients not being virologically suppressed due to missed injections: Somewhat concerned | 0
  Patients not being virologically suppressed due to missed injections: Slightly concerned | 2
  Patients not being virologically suppressed due to missed injections: Not at all concerned | 0
  Patients not being virologically suppressed due to missed injections: Missing | 1
  Being informed (in a timely manner) of adverse events: Extremely concerned | 0
  Being informed (in a timely manner) of adverse events: Moderately concerned | 0
  Being informed (in a timely manner) of adverse events: Somewhat concerned | 0
  Being informed (in a timely manner) of adverse events: Slightly concerned | 1
  Being informed (in a timely manner) of adverse events: Not at all concerned | 1
  Being informed (in a timely manner) of adverse events: Missing | 1
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Extremely concerned | 0
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Moderately concerned | 0
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Somewhat concerned | 1
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Slightly concerned | 0
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Not at all concerned | 1
  IC's ability to address other care needs of patients presenting to CABENUVA appointments: Missing | 1

14. Secondary Outcome: Number of IC/ASA Staff Assessed for Feasibility of CABENUVA Administration in Participants by Other Quantitative Questionnaires Prior to Month 1
Description: The tailored IC staff questionnaire was developed specifically for this study and contains items regarding the staff member's role at the IC, as well as their attitudes, concerns, and anticipated/implemented procedures regarding the use of CABENUVA/long-acting injectable administered by ICs. The IC/ASA staff members were asked to indicate their level of concern across 16 areas of potential concern, on a five-point scale from "not at all concerned" to "extremely concerned."
Time Frame: Prior to Month 1 (Baseline)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 113
Participants
  Understanding how to bridge patients on oral dose for planned missed doses- Extremely concerned | 9
  Understanding how to bridge patients on oral dose for planned missed doses- Moderately concerned | 16
  Understanding how to bridge patients on oral dose for planned missed doses- Somewhat concerned | 17
  Understanding how to bridge patients on oral dose for planned missed doses- Slightly concerned | 37
  Understanding how to bridge patients on oral dose for planned missed doses- Not at all concerned | 33
  Understanding how to bridge patients on oral dose for planned missed doses-Missing | 1
  Management of reporting abnormal lab results with HIV providers- Extremely concerned | 9
  Management of reporting abnormal lab results with HIV providers- Moderately concerned | 11
  Management of reporting abnormal lab results with HIV providers- Somewhat concerned | 15
  Management of reporting abnormal lab results with HIV providers- Slightly concerned | 22
  Management of reporting abnormal lab results with HIV providers- Not at all concerned | 55
  Management of reporting abnormal lab results with HIV providers- Missing | 1
  Understanding when to bridge patients on oral dose for planned missed doses- Extremely concerned | 8
  Understanding when to bridge patients on oral dose for planned missed doses Moderately concerned | 18
  Understanding when to bridge patients on oral dose for planned missed doses Somewhat concerned | 20
  Understanding when to bridge patients on oral dose for planned missed doses- Slightly concerned | 36
  Understanding when to bridge patients on oral dose for planned missed doses Not at all concerned | 30
  Understanding when to bridge patients on oral dose for planned missed doses- Missing | 1
  IC's ability to address other care needs of patients at CABENUVA appointments- Extremely concerned | 6
  IC's ability to address other care needs of patients at CABENUVA appointments- Moderately concerned | 19
  IC's ability to address other care needs of patients at CABENUVA appointments- Somewhat concerned | 20
  IC's ability to address other care needs of patients at CABENUVA appointments- Slightly concerned | 24
  IC's ability to address other care needs of patients at CABENUVA appointments- Not at all concerned | 42
  IC's ability to address other care needs of patients at CABENUVA appointments- Missing | 2
  Frequency of lab draws at the infusion center- Extremely concerned | 6
  Frequency of lab draws at the infusion center- Moderately concerned | 12
  Frequency of lab draws at the infusion center- Somewhat concerned | 23
  Frequency of lab draws at the infusion center- Slightly concerned | 23
  Frequency of lab draws at the infusion center- Not at all concerned | 48
  Frequency of lab draws at the infusion center- Missing | 1
  Management of rescheduling appointments during correct treatment windows- Extremely concerned | 4
  Management of rescheduling appointments during correct treatment windows- Moderately concerned | 5
  Management of rescheduling appointments during correct treatment windows- Somewhat concerned | 8
  Management of rescheduling appointments during correct treatment windows- Slightly concerned | 32
  Management of rescheduling appointments during correct treatment windows- Not at all concerned | 63
  Management of rescheduling appointments during correct treatment windows- Missing | 1
  Management of scheduling appointments during correct treatment windows- Extremely concerned | 4
  Management of scheduling appointments during correct treatment windows- Moderately concerned | 4
  Management of scheduling appointments during correct treatment windows- Somewhat concerned | 10
  Management of scheduling appointments during correct treatment windows- Slightly concerned | 25
  Management of scheduling appointments during correct treatment windows- Not at all concerned | 69
  Management of scheduling appointments during correct treatment windows- Missing | 1
  Answering patient questions between visits- Extremely concerned | 3
  Answering patient questions between visits- Moderately concerned | 10
  Answering patient questions between visits- Somewhat concerned | 18
  Answering patient questions between visits- Slightly concerned | 38
  Answering patient questions between visits- Not at all concerned | 43
  Answering patient questions between visits- Missing | 1
  Management of confirming patient insurance coverage- Extremely concerned | 3
  Management of confirming patient insurance coverage- Moderately concerned | 4
  Management of confirming patient insurance coverage- Somewhat- concerned | 7
  Management of confirming patient insurance coverage- Slightly concerned | 16
  Management of confirming patient insurance coverage- Not at all concerned | 82
  Management of confirming patient insurance coverage- Missing | 1
  Patient insurance coverage clearing for payment- Extremely concerned | 3
  Patient insurance coverage clearing for payment- Moderately concerned | 1
  Patient insurance coverage clearing for payment- Somewhat concerned | 12
  Patient insurance coverage clearing for payment- Slightly concerned | 17
  Patient insurance coverage clearing for payment- Not at all concerned | 79
  Patient insurance coverage clearing for payment- Missing | 1
  Management of patient injection-related pain/soreness- Extremely concerned | 2
  Management of patient injection-related pain/soreness- Moderately concerned | 5
  Management of patient injection-related pain/soreness- Somewhat concerned | 10
  Management of patient injection-related pain/soreness- Slightly concerned | 28
  Management of patient injection-related pain/soreness- Not at all concerned | 67
  Management of patient injection-related pain/soreness- Missing | 1
  Management of reporting of adverse events- Extremely concerned | 2
  Management of reporting of adverse events- Moderately concerned | 4
  Management of reporting of adverse events- Somewhat concerned | 9
  Management of reporting of adverse events- Slightly concerned | 25
  Management of reporting of adverse events- Not at all concerned | 72
  Management of reporting of adverse events- Missing | 1
  Patients' willingness to travel to an infusion center for each injection visit- Extremely concerned | 1
  Patients' willingness to travel to an infusion center for each injection visit- Moderately concerned | 10
  Patients' willingness to travel to an infusion center for each injection visit- Somewhat concerned | 26
  Patients' willingness to travel to an infusion center for each injection visit- Slightly concerned | 14
  Patients' willingness to travel to an infusion center for each injection visit- Not at all concerned | 61
  Patients' willingness to travel to an infusion center for each injection visit- Missing | 1
  Timely reporting of adverse events to HIV providers- Extremely concerned | 0
  Timely reporting of adverse events to HIV providers- Moderately concerned | 5
  Timely reporting of adverse events to HIV providers- Somewhat concerned | 5
  Timely reporting of adverse events to HIV providers- Slightly concerned | 17
  Timely reporting of adverse events to HIV providers- Not at all concerned | 85
  Timely reporting of adverse events to HIV providers- Missing | 1
  Timely reporting to the provider when a patient misses a CABENUVA visit- Extremely concerned | 0
  Timely reporting to the provider when a patient misses a CABENUVA visit- Moderately concerned | 2
  Timely reporting to the provider when a patient misses a CABENUVA visit- Somewhat concerned | 6
  Timely reporting to the provider when a patient misses a CABENUVA visit- Slightly concerned | 21
  Timely reporting to the provider when a patient misses a CABENUVA visit- Not at all concerned | 83
  Timely reporting to the provider when a patient misses a CABENUVA visit- Missing | 1
  Timely reporting to the provider when a patient receives CABENUVA- Extremely concerned | 0
  Timely reporting to the provider when a patient receives CABENUVA- Moderately concerned | 1
  Timely reporting to the provider when a patient receives CABENUVA- Somewhat concerned | 7
  Timely reporting to the provider when a patient receives CABENUVA- Slightly concerned | 16
  Timely reporting to the provider when a patient receives CABENUVA- Not at all concerned | 88
  Timely reporting to the provider when a patient receives CABENUVA- Missing | 1

15. Secondary Outcome: Number of IC/ASA Staff Assessed for Feasibility of CABENUVA Administration in Participants Assessed by Other Quantitative Questionnaires at Month 3
Description: The IC/ASA staff members were asked to indicate their level of concern across 16 areas of potential concern, on a five-point scale from "not at all concerned" to "extremely concerned."
Time Frame: At Month 3
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 38
Participants
  Understanding of how to provide patients with oral medication for planned missed doses: Extremely concerned | 0
  Understanding of how to provide patients with oral medication for planned missed doses: Moderately concerned | 5
  Understanding of how to provide patients with oral medication for planned missed doses: Somewhat concerned | 14
  Understanding of how to provide patients with oral medication for planned missed doses: Slightly concerned | 7
  Understanding of how to provide patients with oral medication for planned missed doses: Not at all concerned | 8
  Understanding of how to provide patients with oral medication for planned missed doses: Missing | 4
  Management of reporting abnormal lab results with HIV providers: Extremely concerned | 1
  Management of reporting abnormal lab results with HIV providers: Moderately concerned | 4
  Management of reporting abnormal lab results with HIV providers: Somewhat concerned | 3
  Management of reporting abnormal lab results with HIV providers: Slightly concerned | 9
  Management of reporting abnormal lab results with HIV providers: Not at all concerned | 17
  Management of reporting abnormal lab results with HIV providers: Missing | 4
  Understanding of when patients should receive oral medication for planned missed doses: Extremely concerned | 1
  Understanding of when patients should receive oral medication for planned missed doses: Moderately concerned | 5
  Understanding of when patients should receive oral medication for planned missed doses: Somewhat concerned | 8
  Understanding of when patients should receive oral medication for planned missed doses: Slightly concerned | 9
  Understanding of when patients should receive oral medication for planned missed doses: Not at all concerned | 11
  Understanding of when patients should receive oral medication for planned missed doses: Missing | 4
  Managing patients presenting to CABENUVA appointments with other care needs to be addressed: Extremely concerned | 2
  Managing patients presenting to CABENUVA appointments with other care needs to be addressed: Moderately concerned | 3
  Managing patients presenting to CABENUVA appointments with other care needs to be addressed: Somewhat concerned | 5
  Managing patients presenting to CABENUVA appointments with other care needs to be addressed: Slightly concerned | 13
  Managing patients presenting to CABENUVA appointments with other care needs to be addressed: Not at all concerned | 11
  Managing patients presenting to CABENUVA appointments with other care needs to be addressed: Missing | 4
  Frequency of lab draws at the infusion center: Extremely concerned | 0
  Frequency of lab draws at the infusion center: Moderately concerned | 4
  Frequency of lab draws at the infusion center: Somewhat concerned | 4
  Frequency of lab draws at the infusion center: Slightly concerned | 14
  Frequency of lab draws at the infusion center: Not at all concerned | 12
  Frequency of lab draws at the infusion center: Missing | 4
  Management of rescheduling appointments during correct treatment windows: Extremely concerned | 0
  Management of rescheduling appointments during correct treatment windows: Moderately concerned | 1
  Management of rescheduling appointments during correct treatment windows: Somewhat concerned | 4
  Management of rescheduling appointments during correct treatment windows: Slightly concerned | 10
  Management of rescheduling appointments during correct treatment windows: Not at all concerned | 19
  Management of rescheduling appointments during correct treatment windows: Missing | 4
  Management of scheduling appointments during correct treatment windows: Extremely concerned | 0
  Management of scheduling appointments during correct treatment windows: Moderately concerned | 0
  Management of scheduling appointments during correct treatment windows: Somewhat concerned | 2
  Management of scheduling appointments during correct treatment windows: Slightly concerned | 7
  Management of scheduling appointments during correct treatment windows: Not at all concerned | 25
  Management of scheduling appointments during correct treatment windows: Missing | 4
  Answering patient questions between visits: Extremely concerned | 1
  Answering patient questions between visits: Moderately concerned | 1
  Answering patient questions between visits: Somewhat concerned | 6
  Answering patient questions between visits: Slightly concerned | 9
  Answering patient questions between visits: Not at all concerned | 17
  Answering patient questions between visits: Missing | 4
  Management of confirming patient insurance coverage: Extremely concerned | 0
  Management of confirming patient insurance coverage: Moderately concerned | 0
  Management of confirming patient insurance coverage: Somewhat concerned | 3
  Management of confirming patient insurance coverage: Slightly concerned | 11
  Management of confirming patient insurance coverage: Not at all concerned | 20
  Management of confirming patient insurance coverage: Missing | 4
  Patient insurance coverage clearing for payment: Extremely concerned | 0
  Patient insurance coverage clearing for payment: Moderately concerned | 0
  Patient insurance coverage clearing for payment: Somewhat concerned | 5
  Patient insurance coverage clearing for payment: Slightly concerned | 9
  Patient insurance coverage clearing for payment: Not at all concerned | 20
  Patient insurance coverage clearing for payment: Missing | 4
  Management of patient injection-related pain/soreness: Extremely concerned | 0
  Management of patient injection-related pain/soreness: Moderately concerned | 2
  Management of patient injection-related pain/soreness: Somewhat concerned | 6
  Management of patient injection-related pain/soreness: Slightly concerned | 7
  Management of patient injection-related pain/soreness: Not at all concerned | 19
  Management of patient injection-related pain/soreness: Missing | 4
  Management of reporting of adverse events: Extremely concerned | 0
  Management of reporting of adverse events: Moderately concerned | 3
  Management of reporting of adverse events: Somewhat concerned | 3
  Management of reporting of adverse events: Slightly concerned | 11
  Management of reporting of adverse events: Not at all concerned | 17
  Management of reporting of adverse events: Missing | 4
  Patients' willingness to travel to an infusion center for each injection visit: Extremely concerned | 0
  Patients' willingness to travel to an infusion center for each injection visit: Moderately concerned | 1
  Patients' willingness to travel to an infusion center for each injection visit: Somewhat concerned | 6
  Patients' willingness to travel to an infusion center for each injection visit: Slightly concerned | 7
  Patients' willingness to travel to an infusion center for each injection visit: Not at all concerned | 20
  Patients' willingness to travel to an infusion center for each injection visit: Missing | 4
  Timely reporting of adverse events to HIV providers: Extremely concerned | 0
  Timely reporting of adverse events to HIV providers: Moderately concerned | 1
  Timely reporting of adverse events to HIV providers: Somewhat concerned | 5
  Timely reporting of adverse events to HIV providers: Slightly concerned | 5
  Timely reporting of adverse events to HIV providers: Not at all concerned | 23
  Timely reporting of adverse events to HIV providers: Missing | 4
  Timely reporting to the provider when a patient misses a CABENUVA visit: Extremely concerned | 0
  Timely reporting to the provider when a patient misses a CABENUVA visit: Moderately concerned | 1
  Timely reporting to the provider when a patient misses a CABENUVA visit: Somewhat concerned | 5
  Timely reporting to the provider when a patient misses a CABENUVA visit: Slightly concerned | 6
  Timely reporting to the provider when a patient misses a CABENUVA visit: Not at all concerned | 22
  Timely reporting to the provider when a patient misses a CABENUVA visit: Missing | 4
  Timely reporting to the provider when a patient receives CABENUVA: Extremely concerned | 0
  Timely reporting to the provider when a patient receives CABENUVA: Moderately concerned | 1
  Timely reporting to the provider when a patient receives CABENUVA: Somewhat concerned | 6
  Timely reporting to the provider when a patient receives CABENUVA: Slightly concerned | 1
  Timely reporting to the provider when a patient receives CABENUVA: Not at all concerned | 26
  Timely reporting to the provider when a patient receives CABENUVA: Missing | 4

16. Secondary Outcome: Number of IC/ASA Staff Assessed for Feasibility of CABENUVA Administration in Participants by Other Quantitative Questionnaires at Month 8
Description: as for outcome 15
Time Frame: At Month 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 26
Participants
  Understanding of how to provide patients with oral medication for planned missed doses: Extremely concerned | 1
  Understanding of how to provide patients with oral medication for planned missed doses: Moderately concerned | 6
  Understanding of how to provide patients with oral medication for planned missed doses: Somewhat concerned | 4
  Understanding of how to provide patients with oral medication for planned missed doses: Slightly concerned | 3
  Understanding of how to provide patients with oral medication for planned missed doses: Not at all concerned | 6
  Understanding of how to provide patients with oral medication for planned missed doses: Missing | 6
  Management of reporting abnormal lab results with HIV providers: Extremely concerned | 0
  Management of reporting abnormal lab results with HIV providers: Moderately concerned | 0
  Management of reporting abnormal lab results with HIV providers: Somewhat concerned | 1
  Management of reporting abnormal lab results with HIV providers: Slightly concerned | 9
  Management of reporting abnormal lab results with HIV providers: Not at all concerned | 10
  Management of reporting abnormal lab results with HIV providers: Missing | 6
  Understanding of when patients should receive oral medication for planned missed doses: Extremely concerned | 1
  Understanding of when patients should receive oral medication for planned missed doses: Moderately concerned | 1
  Understanding of when patients should receive oral medication for planned missed doses: Somewhat concerned | 5
  Understanding of when patients should receive oral medication for planned missed doses: Slightly concerned | 6
  Understanding of when patients should receive oral medication for planned missed doses: Not at all concerned | 7
  Understanding of when patients should receive oral medication for planned missed doses: Missing | 6
  Managing patients presenting to CABENUVA appointments with other care needs to be addressed: Extremely concerned | 1
  Managing patients presenting to CABENUVA appointments with other care needs to be addressed: Moderately concerned | 1
  Managing patients presenting to CABENUVA appointments with other care needs to be addressed: Somewhat concerned | 3
  Managing patients presenting to CABENUVA appointments with other care needs to be addressed: Slightly concerned | 6
  Managing patients presenting to CABENUVA appointments with other care needs to be addressed: Not at all concerned | 9
  Managing patients presenting to CABENUVA appointments with other care needs to be addressed: Missing | 6
  Frequency of lab draws at the infusion center: Extremely concerned | 1
  Frequency of lab draws at the infusion center: Moderately concerned | 1
  Frequency of lab draws at the infusion center: Somewhat concerned | 2
  Frequency of lab draws at the infusion center: Slightly concerned | 7
  Frequency of lab draws at the infusion center: Not at all concerned | 9
  Frequency of lab draws at the infusion center: Missing | 6
  Management of rescheduling appointments during correct treatment windows: Extremely concerned | 0
  Management of rescheduling appointments during correct treatment windows: Moderately concerned | 0
  Management of rescheduling appointments during correct treatment windows: Somewhat concerned | 4
  Management of rescheduling appointments during correct treatment windows: Slightly concerned | 6
  Management of rescheduling appointments during correct treatment windows: Not at all concerned | 10
  Management of rescheduling appointments during correct treatment windows: Missing | 6
  Management of scheduling appointments during correct treatment windows: Extremely concerned | 0
  Management of scheduling appointments during correct treatment windows: Moderately concerned | 0
  Management of scheduling appointments during correct treatment windows: Somewhat concerned | 2
  Management of scheduling appointments during correct treatment windows: Slightly concerned | 8
  Management of scheduling appointments during correct treatment windows: Not at all concerned | 10
  Management of scheduling appointments during correct treatment windows: Missing | 6
  Answering patient questions between visits: Extremely concerned | 0
  Answering patient questions between visits: Moderately concerned | 0
  Answering patient questions between visits: Somewhat concerned | 4
  Answering patient questions between visits: Slightly concerned | 5
  Answering patient questions between visits: Not at all concerned | 11
  Answering patient questions between visits: Missing | 6
  Management of confirming patient insurance coverage: Extremely concerned | 0
  Management of confirming patient insurance coverage: Moderately concerned | 0
  Management of confirming patient insurance coverage: Somewhat concerned | 0
  Management of confirming patient insurance coverage: Slightly concerned | 4
  Management of confirming patient insurance coverage: Not at all concerned | 16
  Management of confirming patient insurance coverage: Missing | 6
  Patient insurance coverage clearing for payment: Extremely concerned | 0
  Patient insurance coverage clearing for payment: Moderately concerned | 0
  Patient insurance coverage clearing for payment: Somewhat concerned | 1
  Patient insurance coverage clearing for payment: Slightly concerned | 5
  Patient insurance coverage clearing for payment: Not at all concerned | 14
  Patient insurance coverage clearing for payment: Missing | 6
  Management of patient injection-related pain/soreness: Extremely concerned | 0
  Management of patient injection-related pain/soreness: Moderately concerned | 0
  Management of patient injection-related pain/soreness: Somewhat concerned | 2
  Management of patient injection-related pain/soreness: Slightly concerned | 5
  Management of patient injection-related pain/soreness: Not at all concerned | 13
  Management of patient injection-related pain/soreness: Missing | 6
  Management of reporting of adverse events: Extremely concerned | 0
  Management of reporting of adverse events: Moderately concerned | 0
  Management of reporting of adverse events: Somewhat concerned | 1
  Management of reporting of adverse events: Slightly concerned | 7
  Management of reporting of adverse events: Not at all concerned | 12
  Management of reporting of adverse events: Missing | 6
  Patients' willingness to travel to an infusion center for each injection visit: Extremely concerned | 0
  Patients' willingness to travel to an infusion center for each injection visit: Moderately concerned | 0
  Patients' willingness to travel to an infusion center for each injection visit: Somewhat concerned | 1
  Patients' willingness to travel to an infusion center for each injection visit: Slightly concerned | 3
  Patients' willingness to travel to an infusion center for each injection visit: Not at all concerned | 15
  Patients' willingness to travel to an infusion center for each injection visit: Missing | 7
  Timely reporting of adverse events to HIV providers: Extremely concerned | 0
  Timely reporting of adverse events to HIV providers: Moderately concerned | 0
  Timely reporting of adverse events to HIV providers: Somewhat concerned | 2
  Timely reporting of adverse events to HIV providers: Slightly concerned | 4
  Timely reporting of adverse events to HIV providers: Not at all concerned | 13
  Timely reporting of adverse events to HIV providers: Missing | 7
  Timely reporting to the provider when a patient misses a CABENUVA visit: Extremely concerned | 0
  Timely reporting to the provider when a patient misses a CABENUVA visit: Moderately concerned | 0
  Timely reporting to the provider when a patient misses a CABENUVA visit: Somewhat concerned | 1
  Timely reporting to the provider when a patient misses a CABENUVA visit: Slightly concerned | 5
  Timely reporting to the provider when a patient misses a CABENUVA visit: Not at all concerned | 13
  Timely reporting to the provider when a patient misses a CABENUVA visit: Missing | 7
  Timely reporting to the provider when a patient receives CABENUVA: Extremely concerned | 0
  Timely reporting to the provider when a patient receives CABENUVA: Moderately concerned | 0
  Timely reporting to the provider when a patient receives CABENUVA: Somewhat concerned | 0
  Timely reporting to the provider when a patient receives CABENUVA: Slightly concerned | 3
  Timely reporting to the provider when a patient receives CABENUVA: Not at all concerned | 16
  Timely reporting to the provider when a patient receives CABENUVA: Missing | 7

17. Secondary Outcome: Number of Participants Assessed for Feasibility of CABENUVA Administration by Qualitative Interviews at Month 8
Description: Qualitative interviews were conducted at Month 8 to evaluate the opinions of participants on the feasibility of CABENUVA administration at IC/ASA.
Time Frame: At Month 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 28
Participants
  Good facilities/environment | 8
  Professional and caring staff | 23
  Consistency of providers | 2
  Protects participants' privacy | 14
  Scheduling flexibility | 4
  Appointment reminders | 1
  Quick and easy administration process | 6
  Hassle-free for participants | 1

18. Secondary Outcome: Number of HIV Care Providers Assessed for Feasibility of CABENUVA Administration in Participants by Qualitative Interviews at Month 8
Description: Qualitative interviews were conducted at Month 8 to evaluate the general opinion of HIV care providers on the feasibility of referring participants to receive CABENUVA at the IC/ASA.
Time Frame: At Month 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- HIV/Care Providers: Eligible HIV Care Providers completed study assessments at each data collection time point.
Arm/Group | HIV/Care Providers
Number analyzed (Participants) | 2
Participants
  Only if insurance requires | 1
  Positive experience thus far | 1

19. Secondary Outcome: Number of IC/ASA Staff Assessed for Feasibility of CABENUVA Administration in Participants by Qualitative Interviews at Month 8
Description: Qualitative interviews were conducted at Month 8 to evaluate the general opinion of IC/ ASA staff on feasibility of CABENUVA administration at the IC/ASA.
Time Frame: At Month 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 12
Participants
  Fits into existing process and practices | 12
  Administration of injection gets easier with experience | 3
  Facilitates implementation | 12
  Scheduling system work arounds to accommodate visit window | 1
  Modifying visit duration to account for all the pieces of administering CABENUVA | 2
  Shortage of private rooms | 4

20. Secondary Outcome: Composite Score of Feasibility Process Indications
Description: Composite score of feasibility process was calculated as the mean of the following four scores: FIM Score, Consent Rate, Show Rate, and Return Rate at Visit, on a 0 to 100 scale, where higher numbers correspond to better feasibility.
Time Frame: Up to and including Month 8
Population: Data was collected at the clinic level and analysis was performed on the Clinics that consented one or more participants for administration of intervention.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Clinics
Groups:
- Clinics: Eligible clinics that consented one or more participants for injection were considered in this arm to evaluate feasibility.
Arm/Group | Clinics
Number analyzed (Participants) | 44
Number analyzed (Clinics) | 14
Scores on a scale | 80.8 (5.46)

21. Secondary Outcome: Change in Composite Score and Each Item of Composite Score Over Time
Description: This outcome measure was planned to evaluate change in composite score from baseline to month 8 according to the protocol. The composite score was however not evaluated as a change over time but as a point in time at month 8 as the components of each of the feasibility composite score (FIM score, consent rate, show rate and return rate) were captured at different time intervals.
Time Frame: Baseline (Month 1) and at Month 8
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Scores on a scale
Units Other Than Participants: Clinics
Arm/Group | Clinics
Number analyzed (Participants) | 44
Number analyzed (Clinics) | 14
Scores on a scale
  FIM score | 84.7 (17.96)
  Consent rate | 52.3 (25.73)
  Show rate | 93.6 (10.49)
  Return rate | 92.7 (13.92)

22. Secondary Outcome: Number of HIV Care Providers Who Agree or Completely Agree (a Score of 4 or Higher) Across All Items on the Acceptability of Intervention Measure (AIM)
Description: AIM was employed to evaluate the acceptability of CABENUVA administration at Infusion Centers/ ASAs. Higher scores for AIM indicate greater acceptability, where each item was scored from 1 to 5: Completely disagree (score=1), disagree (score=2), neither agree or disagree (score=3), agree (score=4), completely agree (score=5).
Time Frame: Months 1 (Baseline), 4, and 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 2
Participants
  At Month 1 (baseline) | 1
  At month 4 | 2
  At month 8 | 1

23. Secondary Outcome: Number of Participants Who Agree or Completely Agree (a Score of 4 or Higher) Across All Items on the AIM
Description: AIM were employed to evaluate the acceptability of CABENUVA administration at Infusion Centers/ ASAs. Higher scores for AIM indicate greater acceptability, where each item was scored from 1 to 5: Completely disagree (score=1), disagree (score=2), neither agree or disagree (score=3), agree (score=4), completely agree (score=5).
Time Frame: Month 1 (Baseline), 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 35
Participants
  At Month 1 (baseline) | 35
  At month 3 | 32
  At month 8 | 33

24. Secondary Outcome: Number of IC/ ASA Staff Who Agree or Completely Agree (a Score of 4 or Higher) Across All Items on the AIM
Description: as for outcome 23
Time Frame: Prior to Month 1 (Baseline), and at Month 3 and 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 47
Participants
  Prior to Month 1 (baseline) | 47
  At month 3 | 13
  At month 8 | 13

25. Secondary Outcome: Change in AIM Score Over Time in HIV Care Providers at Month 4 and 8
Description: The mean score for acceptability of the intervention is calculated by averaging the responses from 4 items. The responses were scored based on a scale of 1 to 5 where 1=completely disagree, 2=disagree, 3=neither agree nor disagree, 4=agree, and 5=completely agree.
Time Frame: Month 1 (Baseline), at Months 4 and 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 3
Scores on a scale
  From baseline to month 4 | 0.33 (0.382)
  From baseline to month 8 | 0.25 (1.414)

26. Secondary Outcome: Change in AIM Score Over Time in Participants at Month 3 and 8
Description: as for outcome 25
Time Frame: Month 1 (Baseline), at Months 3 and 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 36
Scores on a scale
  From baseline to month 3: number analyzed (Participants) | 35
  From baseline to month 3 | 0.03 (0.558)
  From baseline to month 8 | 0.00 (0.604)

27. Secondary Outcome: Change in AIM Score Over Time in IC/ ASA Staff at Month 3 and 8
Description: as for outcome 25
Time Frame: Month 1 (Baseline), at Months 3 and 8
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 34
Scores on a scale
  From baseline to month 3 | -0.24 (0.809)
  From baseline to month 8: number analyzed (Participants) | 20
  From baseline to month 8 | -0.03 (0.778)

28. Secondary Outcome: Number of HIV Care Providers Assessed for Acceptability of CABENUVA Administration in Participants at IC/ ASA by Other Quantitative Questionnaire at Months 1, 4 and 8
Time Frame: At Months 1, 4 and 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 3
Participants
  Month 1- How acceptable was the overall process of interacting with the infusion center so far?: Very acceptable | 1
  Month 1- How acceptable was the overall process of interacting with the infusion center so far?: Somewhat acceptable | 0
  Month 1- How acceptable was the overall process of interacting with the infusion center so far?: A little acceptable | 0
  Month 1- How acceptable was the overall process of interacting with the infusion center so far?: Neutral | 0
  Month 1- How acceptable was the overall process of interacting with the infusion center so far?: A little unacceptable | 1
  Month 1- How acceptable was the overall process of interacting with the infusion center so far?: Somewhat unacceptable | 0
  Month 1- How acceptable was the overall process of interacting with the infusion center so far?: Very unacceptable | 0
  Month 1- How acceptable was the overall process of interacting with the infusion center so far?: I have not interacted with the infusion center yet. | 1
  Month 1- How acceptable was the overall process of interacting with the infusion center so far?: Missing | 0
  Month 4- How acceptable was the overall process of interacting with the infusion center so far?: Very acceptable | 2
  Month 4- How acceptable was the overall process of interacting with the infusion center so far?: Somewhat acceptable | 1
  Month 4- How acceptable was the overall process of interacting with the infusion center so far?: A little acceptable | 0
  Month 4- How acceptable was the overall process of interacting with the infusion center so far?: Neutral | 0
  Month 4- How acceptable was the overall process of interacting with the infusion center so far?: A little unacceptable | 0
  Month 4- How acceptable was the overall process of interacting with the infusion center so far?: Somewhat unacceptable | 0
  Month 4- How acceptable was the overall process of interacting with the infusion center so far?: Very unacceptable | 0
  Month 4- How acceptable was the overall process of interacting with the infusion center so far?: I have not interacted with the infusion center yet. | 0
  Month 4- How acceptable was the overall process of interacting with the infusion center so far?: Missing | 0
  Month 8- How acceptable was the overall process of interacting with the infusion center so far?: Very acceptable | 1
  Month 8- How acceptable was the overall process of interacting with the infusion center so far?: Somewhat acceptable | 1
  Month 8- How acceptable was the overall process of interacting with the infusion center so far?: A little acceptable | 0
  Month 8- How acceptable was the overall process of interacting with the infusion center so far?: Neutral | 0
  Month 8- How acceptable was the overall process of interacting with the infusion center so far?: A little unacceptable | 0
  Month 8- How acceptable was the overall process of interacting with the infusion center so far?: Somewhat unacceptable | 0
  Month 8- How acceptable was the overall process of interacting with the infusion center so far?: Very unacceptable | 0
  Month 8- How acceptable was the overall process of interacting with the infusion center so far?: I have not interacted with the infusion center yet. | 0
  Month 8- How acceptable was the overall process of interacting with the infusion center so far?: Missing | 1

29. Secondary Outcome: Number of Participants Assessed for Acceptability of CABENUVA Administration at IC/ ASA by Other Quantitative Questionnaire in at Months 1, 3 and 8
Description: The participants were asked how acceptable it was to come to the IC/ASA for CABENUVA using a 7-point scale from "very acceptable" to "very unacceptable" where 1= very acceptable, 2= somewhat acceptable, 3= a little acceptable, 4= neutral, 5= a little unacceptable, 6= somewhat unacceptable and 7= very unacceptable.
Time Frame: At Months 1, 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 44
Participants
  Month 1- How acceptable is it to you to come to the infusion center for CABENUVA?: Very acceptable | 34
  Month 1- How acceptable is it to you to come to the infusion center for CABENUVA?: Somewhat acceptable | 6
  Month 1- How acceptable is it to you to come to the infusion center for CABENUVA?: A little acceptable | 0
  Month 1- How acceptable is it to you to come to the infusion center for CABENUVA?: Neutral | 2
  Month 1- How acceptable is it to you to come to the infusion center for CABENUVA?: A little unacceptable | 0
  Month 1- How acceptable is it to you to come to the infusion center for CABENUVA?: Somewhat unacceptable | 1
  Month 1- How acceptable is it to you to come to the infusion center for CABENUVA?: Very unacceptable | 0
  Month 1- How acceptable is it to you to come to the infusion center for CABENUVA?: Missing | 1
  Month 3- How acceptable is it to you to come to the infusion center for CABENUVA?: number analyzed (Participants) | 41
  Month 3- How acceptable is it to you to come to the infusion center for CABENUVA?: Very acceptable | 24
  Month 3- How acceptable is it to you to come to the infusion center for CABENUVA?: Somewhat acceptable | 9
  Month 3- How acceptable is it to you to come to the infusion center for CABENUVA?: A little acceptable | 1
  Month 3- How acceptable is it to you to come to the infusion center for CABENUVA?: Neutral | 0
  Month 3- How acceptable is it to you to come to the infusion center for CABENUVA?: A little unacceptable | 0
  Month 3- How acceptable is it to you to come to the infusion center for CABENUVA?: Somewhat unacceptable | 1
  Month 3- How acceptable is it to you to come to the infusion center for CABENUVA?: Very unacceptable | 1
  Month 3- How acceptable is it to you to come to the infusion center for CABENUVA?: Missing | 5
  Month 8- How acceptable is it to you to come to the infusion center for CABENUVA?: number analyzed (Participants) | 38
  Month 8- How acceptable is it to you to come to the infusion center for CABENUVA?: Very acceptable | 23
  Month 8- How acceptable is it to you to come to the infusion center for CABENUVA?: Somewhat acceptable | 8
  Month 8- How acceptable is it to you to come to the infusion center for CABENUVA?: A little acceptable | 1
  Month 8- How acceptable is it to you to come to the infusion center for CABENUVA?: Neutral | 4
  Month 8- How acceptable is it to you to come to the infusion center for CABENUVA?: A little unacceptable | 0
  Month 8- How acceptable is it to you to come to the infusion center for CABENUVA?: Somewhat unacceptable | 1
  Month 8- How acceptable is it to you to come to the infusion center for CABENUVA?: Very unacceptable | 0
  Month 8- How acceptable is it to you to come to the infusion center for CABENUVA?: Missing | 1

30. Secondary Outcome: Number of IC/ ASA Staff Assessed for Acceptability of CABENUVA Administration in Participants at IC/ ASA by Other Quantitative Questionnaire Prior to Month 1
Time Frame: Prior to Month 1 (Baseline)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 113
Participants
  Extremely concerned | 6
  Moderately concerned | 13
  Somewhat concerned | 22
  Slightly concerned | 21
  Not at all concerned | 51
  Missing | 0

31. Secondary Outcome: Number of IC/ ASA Staff Assessed for Acceptability of CABENUVA Administration in Participants at IC/ ASA by Other Quantitative Questionnaire at Months 3 and 8
Time Frame: At Months 3 and 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 38
Participants
  Month 3- Concern from a personal safety perspective about administering CABENUVA to people with HIV?: Extremely concerned | 0
  Month 3- Concern from a personal safety perspective about administering CABENUVA to people with HIV?: Moderately concerned | 0
  Month 3- Concern from a personal safety perspective about administering CABENUVA to people with HIV?: Somewhat concerned | 5
  Month 3- Concern from a personal safety perspective about administering CABENUVA to people with HIV?: Slightly concerned | 6
  Month 3- Concern from a personal safety perspective about administering CABENUVA to people with HIV?: Not at all concerned | 22
  Month 3- Concern from a personal safety perspective about administering CABENUVA to people with HIV?: Unsure/not applicable to role | 1
  Month 3- Concern from a personal safety perspective about administering CABENUVA to people with HIV?: Missing | 4
  Month 8- Concern from a personal safety perspective about administering CABENUVA to people with HIV?: number analyzed (Participants) | 26
  Month 8- Concern from a personal safety perspective about administering CABENUVA to people with HIV?: Extremely concerned | 0
  Month 8- Concern from a personal safety perspective about administering CABENUVA to people with HIV?: Moderately concerned | 1
  Month 8- Concern from a personal safety perspective about administering CABENUVA to people with HIV?: Somewhat concerned | 3
  Month 8- Concern from a personal safety perspective about administering CABENUVA to people with HIV?: Slightly concerned | 4
  Month 8- Concern from a personal safety perspective about administering CABENUVA to people with HIV?: Not at all concerned | 11
  Month 8- Concern from a personal safety perspective about administering CABENUVA to people with HIV?: Unsure/not applicable to role | 1
  Month 8- Concern from a personal safety perspective about administering CABENUVA to people with HIV?: Missing | 6

32. Secondary Outcome: Number of Participants Assessed for Acceptability of CABENUVA Administration at IC/ASA by Qualitative Interviews at Month 8
Description: Participants were asked about their opinion on acceptability of CABENUVA administration at the IC/ASA.
Time Frame: At Month 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Participants Receiving CABENUVA: Eligible IC/ASA Staff completed study assessments at each data collection time point.
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 28
Participants
  Good facilities/environment | 8
  Professional and caring staff | 23
  Consistency of providers | 2
  Protects participants' privacy | 14
  Scheduling flexibility | 4
  Appointment reminders | 1
  Quick and easy administration process | 6
  Hassle-free for participants | 1

33. Secondary Outcome: Number of HIV Care Providers Assessed for Acceptability of CABENUVA Administration in Participants at IC/ASA by Qualitative Interviews at Month 8
Description: HIV care providers were asked about their opinion on the acceptability of participants receiving CABENUVA at the IC/ASA.
Time Frame: At Month 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 2
Participants | 2

34. Secondary Outcome: Number of IC/ASA Staff Assessed for Acceptability of CABENUVA Administration in Participants at IC/ASA by Qualitative Interviews at Month 8
Description: IC/ASA staff were asked about their opinion on the acceptability of administering CABENUVA at an IC/ASA.
Time Frame: At Month 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 12
Participants
  Learned more about CABENUVA | 2
  Improved outlook about CABENUVA | 1
  Ease of administration over time | 2
  Quick and easy administration process | 4
  Easy to integrate into IC/ASA workflow | 4

35. Secondary Outcome: Number of Expert Panel That Agree or Completely Agree (a Score of 4 or Higher) Across All Items on the FIM Scale
Time Frame: Prior to Month 1 (Baseline), and at Month 3 and 6
Population: Analysis was performed on the Expert Panel which includes any Expert Panel member who completed any portion of any questionnaire at the specified timepoint.
Measure: Count of Participants; unit: Participants
Groups:
- Expert Panel: Pre-determined Expert Panel comprising of selected HIV care providers and key IC staff completed study assessments at each data collection time point.
Arm/Group | Expert Panel
Number analyzed (Participants) | 8
Participants
  Prior to Month 1 (Baseline) | 5
  Month 3 | 5
  Month 6 | 5

36. Secondary Outcome: Number of Expert Panel That Agree or Completely Agree (a Score of 4 or Higher) Across All Items on the AIM Scale
Time Frame: Prior to Month 1 (Baseline), and at Month 3 and 6
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Expert Panel
Number analyzed (Participants) | 8
Participants
  Prior to Month 1 (Baseline) | 6
  Month 3 | 6
  Month 6 | 6

37. Secondary Outcome: Change in FIM Score of Expert Panel Over Time Through Month 6
Time Frame: Prior to Month 1 (Baseline) and Up to Month 6
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Expert Panel
Number analyzed (Participants) | 8
Scores on a scale
  Prior to Month 1 (Baseline) | 4.00 (0.991)
  Month 6 | 4.46 (0.534)

38. Secondary Outcome: Change in AIM Score of Expert Panel Over Time Through Month 6
Time Frame: Prior to Month 1 (Baseline) and Up to Month 6
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Expert Panel
Number analyzed (Participants) | 8
Scores on a scale
  Prior to Month 1 (Baseline) | 4.22 (0.619)
  Month 6 | 4.46 (0.510)

39. Secondary Outcome: Number of Expert Panel Members Assessed for Feasibility, Acceptability and Process of Insurance Coverage for CABENUVA Administration in Participants by Quantitative Questionnaires Prior to Month 1
Time Frame: Prior to Month 1 (Baseline)
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Expert Panel
Number analyzed (Participants) | 8
Participants
  What is your preference for who will conduct the insurance benefit verification?: Infusion Center Staff | 4
  What is your preference for who will conduct the insurance benefit verification?: Unsure/Not applicable to role | 2
  What is your preference for who will conduct the insurance benefit verification?: HIV Provider/ Clinic Staff | 1
  What is your preference for who will conduct the insurance benefit verification?: ViiV Connect (reimbursement hub) | 1
  What is your preference for who will conduct the insurance benefit verification?: Missing | 0
  What is your preference for who notifies the patient about insurance coverage?: Infusion Center Staff | 6
  What is your preference for who notifies the patient about insurance coverage?: Unsure/Not applicable to role | 2
  What is your preference for who notifies the patient about insurance coverage?: HIV Provider/ Clinic Staff | 2
  What is your preference for who notifies the patient about insurance coverage?: ViiV Connect (reimbursement hub) | NA — This category is not applicable to this question.
  What is your preference for who notifies the patient about insurance coverage?: Missing | 0

40. Secondary Outcome: Number of Expert Panel Members Assessed for Feasibility, Acceptability and Process of Communication for CABENUVA Administration in Participants by Quantitative Questionnaires Prior to Month 1
Time Frame: Prior to Month 1 (Baseline)
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Expert Panel
Number analyzed (Participants) | 8
Participants
  Preferred mode of communication between HIV provider and IC when a patient discontinues CABENUVA: Fax | 5
  Preferred mode of communication between HIV provider and IC when a patient discontinues CABENUVA: Phone call | 2
  Preferred mode of communication between HIV provider and IC when a patient discontinues CABENUVA: Secure Electronic Medical Record message | 1
  Preferred mode of communication between HIV provider and IC when a patient discontinues CABENUVA: Text | 0
  Preferred mode of communication between HIV provider and IC when a patient discontinues CABENUVA: Email | 0
  Preferred mode of communication between HIV provider and IC when a patient discontinues CABENUVA: Other | 0
  Preferred mode of communication between HIV provider and IC when a patient discontinues CABENUVA: Unsure/ Not applicable to role | 0
  Preferred mode of communication between HIV provider and IC when a patient discontinues CABENUVA: Missing | 0
  Preferred mode of communication about AEs from IC to HIV provider: Fax | 5
  Preferred mode of communication about AEs from IC to HIV provider: Phone call | 2
  Preferred mode of communication about AEs from IC to HIV provider: Secure Electronic Medical Record message | 1
  Preferred mode of communication about AEs from IC to HIV provider: Text | 0
  Preferred mode of communication about AEs from IC to HIV provider: Email | 0
  Preferred mode of communication about AEs from IC to HIV provider: Other | 0
  Preferred mode of communication about AEs from IC to HIV provider: Unsure/ Not applicable to role | 0
  Preferred mode of communication about AEs from IC to HIV provider: Missing | 0

41. Secondary Outcome: Number of Expert Panel Members Assessed for Feasibility, Acceptability and Process of CABENUVA Administration (Interval of Time) in Participants by Quantitative Questionnaires Prior to Month 1
Description: In this outcome measure, Expert Panel members were asked about their views on the IC/ASA administration model (for patients receiving CABENUVA injections at the infusion center, what is the preferred interval of time for patients to be seen by their HIV provider).
Time Frame: Prior to Month 1 (Baseline)
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Expert Panel
Number analyzed (Participants) | 8
Participants
  Never/ not needed | 0
  Every month | 0
  Every 2 months | 0
  Every 3 months | 1
  Every 4 months | 1
  Every 6 months | 2
  Yearly | 2
  As needed (i.e., when an adverse event occurs) | 1
  Unsure/ Not applicable to role | 2
  Missing | 0

42. Secondary Outcome: Number of Expert Panel Members Assessed for Feasibility, Acceptability and Process of Referring Participants for CABENUVA Administration by Quantitative Questionnaires Prior to Month 1
Time Frame: Prior to Month 1 (Baseline)
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Expert Panel
Number analyzed (Participants) | 8
Participants
  Fax | 5
  Unsure/Not applicable to role | 2
  Secure Electronic Medical Record message | 1
  Phone call | 0
  Email | 0
  Other | 0
  Missing | 0

43. Secondary Outcome: Number of Expert Panel Members Assessed for Feasibility, Acceptability and Process of Insurance and Communication for CABENUVA Administration in Participants by Quantitative Questionnaires at Month 3
Time Frame: At Month 3
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Expert Panel
Number analyzed (Participants) | 7
Participants
  Acceptability of insurance verification/confirmation process for patients referred to the IC: number analyzed (Participants) | 3
  Acceptability of insurance verification/confirmation process for patients referred to the IC: Extremely acceptable | 0
  Acceptability of insurance verification/confirmation process for patients referred to the IC: Very acceptable | 0
  Acceptability of insurance verification/confirmation process for patients referred to the IC: Somewhat acceptable | 1
  Acceptability of insurance verification/confirmation process for patients referred to the IC: Neither acceptable nor unacceptable | 0
  Acceptability of insurance verification/confirmation process for patients referred to the IC: Somewhat unacceptable | 0
  Acceptability of insurance verification/confirmation process for patients referred to the IC: Very unacceptable | 1
  Acceptability of insurance verification/confirmation process for patients referred to the IC: Extremely unacceptable | 0
  Acceptability of insurance verification/confirmation process for patients referred to the IC: I do not have knowledge of/not involved in this process | 1
  How acceptable has the process been for relaying insurance coverage information to patients?: number analyzed (Participants) | 3
  How acceptable has the process been for relaying insurance coverage information to patients?: Extremely acceptable | 1
  How acceptable has the process been for relaying insurance coverage information to patients?: Very acceptable | 1
  How acceptable has the process been for relaying insurance coverage information to patients?: Somewhat acceptable | 0
  How acceptable has the process been for relaying insurance coverage information to patients?: Neither acceptable nor unacceptable | 0
  How acceptable has the process been for relaying insurance coverage information to patients?: Somewhat unacceptable | 1
  How acceptable has the process been for relaying insurance coverage information to patients?: Very unacceptable | 0
  How acceptable has the process been for relaying insurance coverage information to patients?: Extremely unacceptable | 0
  How acceptable has the process been for relaying insurance coverage information to patients?: I do not have knowledge of/not involved in this process | 0
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: Extremely acceptable | 0
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: Very acceptable | 1
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: Somewhat acceptable | 1
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: Neither acceptable nor unacceptable | 1
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: Somewhat unacceptable | 1
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: Very unacceptable | 0
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: Extremely unacceptable | 0
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: I do not have knowledge of/not involved in this process | 3

44. Secondary Outcome: Number of Expert Panel Members Assessed for Feasibility, Acceptability and Process of Insurance and Communication for CABENUVA Administration in Participants by Quantitative Questionnaires at Month 6
Time Frame: At Month 6
Population: as for outcome 35
Measure: Count of Participants; unit: Participants
Arm/Group | Expert Panel
Number analyzed (Participants) | 6
Participants
  Acceptability of insurance verification/confirmation process for patients referred to the IC: number analyzed (Participants) | 2
  Acceptability of insurance verification/confirmation process for patients referred to the IC: Extremely acceptable | 0
  Acceptability of insurance verification/confirmation process for patients referred to the IC: Very acceptable | 0
  Acceptability of insurance verification/confirmation process for patients referred to the IC: Somewhat acceptable | 1
  Acceptability of insurance verification/confirmation process for patients referred to the IC: Neither acceptable nor unacceptable | 0
  Acceptability of insurance verification/confirmation process for patients referred to the IC: Somewhat unacceptable | 0
  Acceptability of insurance verification/confirmation process for patients referred to the IC: Very unacceptable | 0
  Acceptability of insurance verification/confirmation process for patients referred to the IC: Extremely unacceptable | 0
  Acceptability of insurance verification/confirmation process for patients referred to the IC: I do not have knowledge of/not involved in this process | 1
  How acceptable has the process been for relaying insurance coverage information to patients?: number analyzed (Participants) | 1
  How acceptable has the process been for relaying insurance coverage information to patients?: Extremely acceptable | 0
  How acceptable has the process been for relaying insurance coverage information to patients?: Very acceptable | 1
  How acceptable has the process been for relaying insurance coverage information to patients?: Somewhat acceptable | 0
  How acceptable has the process been for relaying insurance coverage information to patients?: Neither acceptable nor unacceptable | 0
  How acceptable has the process been for relaying insurance coverage information to patients?: Somewhat unacceptable | 0
  How acceptable has the process been for relaying insurance coverage information to patients?: Very unacceptable | 0
  How acceptable has the process been for relaying insurance coverage information to patients?: Extremely unacceptable | 0
  How acceptable has the process been for relaying insurance coverage information to patients?: I do not have knowledge of/not involved in this process | 0
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: Extremely acceptable | 0
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: Very acceptable | 1
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: Somewhat acceptable | 1
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: Neither acceptable nor unacceptable | 0
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: Somewhat unacceptable | 0
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: Very unacceptable | 0
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: Extremely unacceptable | 0
  Acceptability of communication between yourself and the IC during the oral lead-in phase?: I do not have knowledge of/not involved in this process | 4

45. Secondary Outcome: Number of Expert Panel Members Assessed for Feasibility, Acceptability and Process of CABENUVA Administration in Participants by Qualitative Interviews Prior to Month 1
Description: The Expert Panel were asked about the key steps focused on the process of CABENUVA administration at IC/ASAs in order to inform the development of the blueprint.
Time Frame: Prior to Month 1 (Baseline)
Population: Analysis was performed on the Expert Panel which includes any Expert Panel member who completed any portion of any questionnaire at the specified timepoint study.
Measure: Count of Participants; unit: Participants
Arm/Group | Expert Panel
Number analyzed (Participants) | 8
Participants
  Staff Identify patients for CABENUVA and discuss with patient | 2
  Staff formally refer patients to verify insurance | 4
  Staff initiates patient on oral lead-in | 3
  Staff schedules first patient visit and conducts pre-visit steps | 2
  Patient attends first injection appointment | 1
  Post injection reporting and future appointment scheduling | 2

46. Secondary Outcome: Number of Expert Panel Members Assessed for Feasibility, Acceptability and Process of CABENUVA Administration in Participants by Qualitative Interviews at Month 6
Description: as for outcome 45
Time Frame: At Month 6
Population: as for outcome 45
Measure: Count of Participants; unit: Participants
Arm/Group | Expert Panel
Number analyzed (Participants) | 8
Participants
  Staff Identify patients for CABENUVA and discuss with patient | 2
  Staff formally refer patients to verify insurance | 3
  Staff initiates patient on oral lead-in | 2
  Staff schedules first patient visit and conducts pre-visit steps | 1
  Patient attends first injection appointment | 4
  Post injection reporting and future appointment scheduling | 5

47. Secondary Outcome: Number of Participants Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration With Other Quantitative Questionnaires at Month 1
Time Frame: At Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 44
Participants
  Concern about unwanted disclosure of HIV status when attending appointments at HIV providers office: Very concerned | 12
  Concern about unwanted disclosure of HIV status when attending appointments at HIV providers office: Moderately concerned | 7
  Concern about unwanted disclosure of HIV status when attending appointments at HIV providers office: Somewhat concerned | 4
  Concern about unwanted disclosure of HIV status when attending appointments at HIV providers office: A little concerned | 3
  Concern about unwanted disclosure of HIV status when attending appointments at HIV providers office: Not at all concerned | 17
  Concern about unwanted disclosure of HIV status when attending appointments at HIV providers office: Missing | 1
  Concern about unwanted disclosure of HIV status when attending appointments at IC: Very concerned | 10
  Concern about unwanted disclosure of HIV status when attending appointments at IC: Moderately concerned | 5
  Concern about unwanted disclosure of HIV status when attending appointments at IC: Somewhat concerned | 5
  Concern about unwanted disclosure of HIV status when attending appointments at IC: A little concerned | 5
  Concern about unwanted disclosure of HIV status when attending appointments at IC: Not at all concerned | 18
  Concern about unwanted disclosure of HIV status when attending appointments at IC: Missing | 1

48. Secondary Outcome: Number of Participants Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration With Other Quantitative Questionnaires (Q 1) at Month 3 and 8
Time Frame: At Month 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 41
Participants
  Month 3- Have you been treated differently, or experienced stigma or discrimination at the IC?: Yes | 1
  Month 3- Have you been treated differently, or experienced stigma or discrimination at the IC?: No | 34
  Month 3- Have you been treated differently, or experienced stigma or discrimination at the IC?: Prefer not to answer | 1
  Month 3- Have you been treated differently, or experienced stigma or discrimination at the IC?: Missing | 5
  Month 8- Have you been treated differently, or experienced stigma or discrimination at the IC?: number analyzed (Participants) | 38
  Month 8- Have you been treated differently, or experienced stigma or discrimination at the IC?: Yes | 1
  Month 8- Have you been treated differently, or experienced stigma or discrimination at the IC?: No | 34
  Month 8- Have you been treated differently, or experienced stigma or discrimination at the IC?: Prefer not to answer | 2
  Month 8- Have you been treated differently, or experienced stigma or discrimination at the IC?: Missing | 1

49. Secondary Outcome: Number of Participants Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration With Other Quantitative Questionnaires (Q 2) at Months 3 and 8
Time Frame: At Months 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 1
Participants
  Month 3- Your experience at IC compared to your experience at your HIV provider's office/clinic?: A lot worse | 0
  Month 3- Your experience at IC compared to your experience at your HIV provider's office/clinic?: Somewhat worse | 0
  Month 3- Your experience at IC compared to your experience at your HIV provider's office/clinic?: A little worse | 0
  Month 3- Your experience at IC compared to your experience at your HIV provider's office/clinic?: About the same | 1
  Month 3- Your experience at IC compared to your experience at your HIV provider's office/clinic?: A little better | 0
  Month 3- Your experience at IC compared to your experience at your HIV provider's office/clinic?: Somewhat better | 0
  Month 3- Your experience at IC compared to your experience at your HIV provider's office/clinic?: A lot better | 0
  Month 8- Your experience at IC compared to your experience at your HIV provider's office/clinic?: A lot worse | 0
  Month 8- Your experience at IC compared to your experience at your HIV provider's office/clinic?: Somewhat worse | 0
  Month 8- Your experience at IC compared to your experience at your HIV provider's office/clinic?: A little worse | 1
  Month 8- Your experience at IC compared to your experience at your HIV provider's office/clinic?: About the same | 0
  Month 8- Your experience at IC compared to your experience at your HIV provider's office/clinic?: A little better | 0
  Month 8- Your experience at IC compared to your experience at your HIV provider's office/clinic?: Somewhat better | 0
  Month 8- Your experience at IC compared to your experience at your HIV provider's office/clinic?: A lot better | 0

50. Secondary Outcome: Number of Participants Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration With Other Quantitative Questionnaires (Q 3) at Months 3 and 8
Time Frame: At Months 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 1
Participants
  Month 3- Do you believe you have been treated differently based on any of the following factors.: Age | 0
  Month 3- Do you believe you have been treated differently based on any of the following factors.: Race/ethnicity | 0
  Month 3- Do you believe you have been treated differently based on any of the following factors.: Sex | 0
  Month 3- Do you believe you have been treated differently based on any of the following factors.: Gender identity | 0
  Month 3- Do you believe you have been treated differently based on any of the following factors.: Sexual preference | 0
  Month 3- Do you believe you have been treated differently based on any of the following factors.: HIV status | 0
  Month 3- Do you believe you have been treated differently based on any of the following factors.: Religion | 0
  Month 3- Do you believe you have been treated differently based on any of the following factors.: Physical appearance | 0
  Month 3- Do you believe you have been treated differently based on any of the following factors.: Housing status | 0
  Month 3- Do you believe you have been treated differently based on any of the following factors.: Due to pregnancy/being pregnant | 0
  Month 3- Do you believe you have been treated differently based on any of the following factors.: Other | 0
  Month 3- Do you believe you have been treated differently based on any of the following factors.: None of the above | 1
  Month 8- Do you believe you have been treated differently based on any of the following factors.: Age | 0
  Month 8- Do you believe you have been treated differently based on any of the following factors.: Race/ethnicity | 0
  Month 8- Do you believe you have been treated differently based on any of the following factors.: Sex | 0
  Month 8- Do you believe you have been treated differently based on any of the following factors.: Gender identity | 0
  Month 8- Do you believe you have been treated differently based on any of the following factors.: Sexual preference | 0
  Month 8- Do you believe you have been treated differently based on any of the following factors.: HIV status | 0
  Month 8- Do you believe you have been treated differently based on any of the following factors.: Religion | 0
  Month 8- Do you believe you have been treated differently based on any of the following factors.: Physical appearance | 0
  Month 8- Do you believe you have been treated differently based on any of the following factors.: Housing status | 0
  Month 8- Do you believe you have been treated differently based on any of the following factors.: Due to pregnancy/being pregnant | 0
  Month 8- Do you believe you have been treated differently based on any of the following factors.: Other | 0
  Month 8- Do you believe you have been treated differently based on any of the following factors.: None of the above | 1

51. Secondary Outcome: Number of Participants Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration With Other Quantitative Questionnaires (Q 4) at Months 3 and 8
Time Frame: At Months 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 41
Participants
  Month 3- How comfortable are you with the infusion center managing your CABENUVA injections?: Extremely comfortable | 28
  Month 3- How comfortable are you with the infusion center managing your CABENUVA injections?: Very comfortable | 6
  Month 3- How comfortable are you with the infusion center managing your CABENUVA injections?: Somewhat comfortable | 2
  Month 3- How comfortable are you with the infusion center managing your CABENUVA injections?: Neutral | 0
  Month 3- How comfortable are you with the infusion center managing your CABENUVA injections?: Somewhat uncomfortable | 0
  Month 3- How comfortable are you with the infusion center managing your CABENUVA injections?: Very uncomfortable | 0
  Month 3- How comfortable are you with the infusion center managing your CABENUVA injections?: Extremely uncomfortable | 0
  Month 3- How comfortable are you with the infusion center managing your CABENUVA injections?: Missing | 5
  Month 8- How comfortable are you with the infusion center managing your CABENUVA injections?: number analyzed (Participants) | 38
  Month 8- How comfortable are you with the infusion center managing your CABENUVA injections?: Extremely comfortable | 24
  Month 8- How comfortable are you with the infusion center managing your CABENUVA injections?: Very comfortable | 10
  Month 8- How comfortable are you with the infusion center managing your CABENUVA injections?: Somewhat comfortable | 1
  Month 8- How comfortable are you with the infusion center managing your CABENUVA injections?: Neutral | 0
  Month 8- How comfortable are you with the infusion center managing your CABENUVA injections?: Somewhat uncomfortable | 1
  Month 8- How comfortable are you with the infusion center managing your CABENUVA injections?: Very uncomfortable | 0
  Month 8- How comfortable are you with the infusion center managing your CABENUVA injections?: Extremely uncomfortable | 0
  Month 8- How comfortable are you with the infusion center managing your CABENUVA injections?: Missing | 2

52. Secondary Outcome: Number of Participants Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration With Other Quantitative Questionnaires (Q 5) at Months 3 and 8
Time Frame: At Months 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 41
Participants
  Month 3- How welcome do you feel at the infusion center?: Extremely welcome | 25
  Month 3- How welcome do you feel at the infusion center?: Very welcome | 10
  Month 3- How welcome do you feel at the infusion center?: Somewhat welcome | 0
  Month 3- How welcome do you feel at the infusion center?: Neutral | 1
  Month 3- How welcome do you feel at the infusion center?: Somewhat unwelcome | 0
  Month 3- How welcome do you feel at the infusion center?: Very unwelcome | 0
  Month 3- How welcome do you feel at the infusion center?: Extremely unwelcome | 0
  Month 3- How welcome do you feel at the infusion center?: Missing | 5
  Month 8- How welcome do you feel at the infusion center?: number analyzed (Participants) | 38
  Month 8- How welcome do you feel at the infusion center?: Extremely welcome | 29
  Month 8- How welcome do you feel at the infusion center?: Very welcome | 7
  Month 8- How welcome do you feel at the infusion center?: Somewhat welcome | 0
  Month 8- How welcome do you feel at the infusion center?: Neutral | 1
  Month 8- How welcome do you feel at the infusion center?: Somewhat unwelcome | 0
  Month 8- How welcome do you feel at the infusion center?: Very unwelcome | 0
  Month 8- How welcome do you feel at the infusion center?: Extremely unwelcome | 0
  Month 8- How welcome do you feel at the infusion center?: Missing | 1

53. Secondary Outcome: Number of Participants Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration With Other Quantitative Questionnaires (Q 6) at Months 3 and 8
Time Frame: At Months 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 41
Participants
  Month 3- How respectful are the infusion center staff when you are there for your injections?: Extremely respectful | 30
  Month 3- How respectful are the infusion center staff when you are there for your injections?: Very respectful | 6
  Month 3- How respectful are the infusion center staff when you are there for your injections?: Somewhat respectful | 0
  Month 3- How respectful are the infusion center staff when you are there for your injections?: Neutral | 0
  Month 3- How respectful are the infusion center staff when you are there for your injections?: Somewhat unrespectful | 0
  Month 3- How respectful are the infusion center staff when you are there for your injections?: Very unrespectful | 0
  Month 3- How respectful are the infusion center staff when you are there for your injections?: Extremely unrespectful | 0
  Month 3- How respectful are the infusion center staff when you are there for your injections?: Missing | 5
  Month 8- How respectful are the infusion center staff when you are there for your injections?: number analyzed (Participants) | 38
  Month 8- How respectful are the infusion center staff when you are there for your injections?: Extremely respectful | 31
  Month 8- How respectful are the infusion center staff when you are there for your injections?: Very respectful | 6
  Month 8- How respectful are the infusion center staff when you are there for your injections?: Somewhat respectful | 0
  Month 8- How respectful are the infusion center staff when you are there for your injections?: Neutral | 0
  Month 8- How respectful are the infusion center staff when you are there for your injections?: Somewhat unrespectful | 0
  Month 8- How respectful are the infusion center staff when you are there for your injections?: Very unrespectful | 0
  Month 8- How respectful are the infusion center staff when you are there for your injections?: Extremely unrespectful | 0
  Month 8- How respectful are the infusion center staff when you are there for your injections?: Missing | 1

54. Secondary Outcome: Number of Participants Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration With Other Quantitative Questionnaires (Q 7) at Months 3 and 8
Time Frame: At Months 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 41
Participants
  Month 3- Satisfaction level of privacy at the IC for receiving your injections?: Extremely satisfied | 25
  Month 3- Satisfaction level of privacy at the IC for receiving your injections?: Very satisfied | 9
  Month 3- Satisfaction level of privacy at the IC for receiving your injections?: Somewhat satisfied | 1
  Month 3- Satisfaction level of privacy at the IC for receiving your injections?: Neutral | 1
  Month 3- Satisfaction level of privacy at the IC for receiving your injections?: Somewhat dissatisfied | 0
  Month 3- Satisfaction level of privacy at the IC for receiving your injections?: Very dissatisfied | 0
  Month 3- Satisfaction level of privacy at the IC for receiving your injections?: Extremely dissatisfied | 0
  Month 3- Satisfaction level of privacy at the IC for receiving your injections?: Missing | 5
  Month 8- Satisfaction level of privacy at the IC for receiving your injections?: number analyzed (Participants) | 38
  Month 8- Satisfaction level of privacy at the IC for receiving your injections?: Extremely satisfied | 27
  Month 8- Satisfaction level of privacy at the IC for receiving your injections?: Very satisfied | 6
  Month 8- Satisfaction level of privacy at the IC for receiving your injections?: Somewhat satisfied | 1
  Month 8- Satisfaction level of privacy at the IC for receiving your injections?: Neutral | 1
  Month 8- Satisfaction level of privacy at the IC for receiving your injections?: Somewhat dissatisfied | 1
  Month 8- Satisfaction level of privacy at the IC for receiving your injections?: Very dissatisfied | 1
  Month 8- Satisfaction level of privacy at the IC for receiving your injections?: Extremely dissatisfied | 0
  Month 8- Satisfaction level of privacy at the IC for receiving your injections?: Missing | 1

55. Secondary Outcome: Number of Participants Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration With Other Quantitative Questionnaires (Q 8) at Months 3 and 8
Time Frame: At Months 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 41
Participants
  Month 3- How convenient is it for you to get to the infusion center for your CABENUVA visits?: Very convenient | 20
  Month 3- How convenient is it for you to get to the infusion center for your CABENUVA visits?: Somewhat convenient | 7
  Month 3- How convenient is it for you to get to the infusion center for your CABENUVA visits?: A little convenient | 3
  Month 3- How convenient is it for you to get to the infusion center for your CABENUVA visits?: Neutral | 1
  Month 3- How convenient is it for you to get to the infusion center for your CABENUVA visits?: A little inconvenient | 2
  Month 3- How convenient is it for you to get to the infusion center for your CABENUVA visits?: Somewhat inconvenient | 3
  Month 3- How convenient is it for you to get to the infusion center for your CABENUVA visits?: Very inconvenient | 0
  Month 3- How convenient is it for you to get to the infusion center for your CABENUVA visits?: Missing | 5
  Month 8- How convenient is it for you to get to the infusion center for your CABENUVA visits?: number analyzed (Participants) | 38
  Month 8- How convenient is it for you to get to the infusion center for your CABENUVA visits?: Very convenient | 23
  Month 8- How convenient is it for you to get to the infusion center for your CABENUVA visits?: Somewhat convenient | 4
  Month 8- How convenient is it for you to get to the infusion center for your CABENUVA visits?: A little convenient | 3
  Month 8- How convenient is it for you to get to the infusion center for your CABENUVA visits?: Neutral | 3
  Month 8- How convenient is it for you to get to the infusion center for your CABENUVA visits?: A little inconvenient | 2
  Month 8- How convenient is it for you to get to the infusion center for your CABENUVA visits?: Somewhat inconvenient | 1
  Month 8- How convenient is it for you to get to the infusion center for your CABENUVA visits?: Very inconvenient | 1
  Month 8- How convenient is it for you to get to the infusion center for your CABENUVA visits?: Missing | 1

56. Secondary Outcome: Number of Participants Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration With Other Quantitative Questionnaires (Q 9) at Months 3 and 8
Time Frame: At Months 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 41
Participants
  Month 3- How long does it typically take you to get to the infusion center?: 1-15 minutes | 9
  Month 3- How long does it typically take you to get to the infusion center?: 16-30 minutes | 12
  Month 3- How long does it typically take you to get to the infusion center?: 31-45 minutes | 9
  Month 3- How long does it typically take you to get to the infusion center?: 46-60 minutes | 5
  Month 3- How long does it typically take you to get to the infusion center?: More than 60 minutes | 0
  Month 3- How long does it typically take you to get to the infusion center?: Missing | 6
  Month 8- How long does it typically take you to get to the infusion center?: number analyzed (Participants) | 38
  Month 8- How long does it typically take you to get to the infusion center?: 1-15 minutes | 8
  Month 8- How long does it typically take you to get to the infusion center?: 16-30 minutes | 15
  Month 8- How long does it typically take you to get to the infusion center?: 31-45 minutes | 11
  Month 8- How long does it typically take you to get to the infusion center?: 46-60 minutes | 1
  Month 8- How long does it typically take you to get to the infusion center?: More than 60 minutes | 2
  Month 8- How long does it typically take you to get to the infusion center?: Missing | 1

57. Secondary Outcome: Number of Participants Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration With Other Quantitative Questionnaires (Q 10) at Months 3 and 8
Description: Participants were asked their opinion on who did they reach out to obtain answers to their questions.
Time Frame: At Months 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 41
Participants
  Month 3- My regular HIV provider | 18
  Month 3- Staff at infusion center | 15
  Month 3- No questions to date | 9
  Month 3- Other staff at my regular HIV provider's office | 0
  Month 3- Other people with HIV | 0
  Month 3- Social media | 0
  Month 3- Missing | 5
  Month 8- My regular HIV provider: number analyzed (Participants) | 38
  Month 8- My regular HIV provider | 20
  Month 8- Staff at the infusion center: number analyzed (Participants) | 38
  Month 8- Staff at the infusion center | 18
  Month 8- No questions to date: number analyzed (Participants) | 38
  Month 8- No questions to date | 11
  Month 8- Other staff at my regular HIV provider's office: number analyzed (Participants) | 38
  Month 8- Other staff at my regular HIV provider's office | 2
  Month 8- Other people with HIV: number analyzed (Participants) | 38
  Month 8- Other people with HIV | 1
  Month 8- Social media: number analyzed (Participants) | 38
  Month 8- Social media | 1
  Month 8- Missing: number analyzed (Participants) | 38
  Month 8- Missing | 1

58. Secondary Outcome: Number of Participants Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration With Other Quantitative Questionnaires (Q 11) at Months 3 and 8
Time Frame: At Months 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 41
Participants
  Month 3- Concern about unwanted disclosure of HIV status when attending appointments at the IC?: Very concerned | 2
  Month 3- Concern about unwanted disclosure of HIV status when attending appointments at the IC?: Moderately concerned | 5
  Month 3- Concern about unwanted disclosure of HIV status when attending appointments at the IC?: Somewhat concerned | 6
  Month 3- Concern about unwanted disclosure of HIV status when attending appointments at the IC?: A little concerned | 1
  Month 3- Concern about unwanted disclosure of HIV status when attending appointments at the IC?: Not at all concerned | 22
  Month 3- Concern about unwanted disclosure of HIV status when attending appointments at the IC?: Missing | 5
  Month 8- Concern about unwanted disclosure of HIV status when attending appointments at the IC?: number analyzed (Participants) | 38
  Month 8- Concern about unwanted disclosure of HIV status when attending appointments at the IC?: Very concerned | 5
  Month 8- Concern about unwanted disclosure of HIV status when attending appointments at the IC?: Moderately concerned | 1
  Month 8- Concern about unwanted disclosure of HIV status when attending appointments at the IC?: Somewhat concerned | 4
  Month 8- Concern about unwanted disclosure of HIV status when attending appointments at the IC?: A little concerned | 5
  Month 8- Concern about unwanted disclosure of HIV status when attending appointments at the IC?: Not at all concerned | 22
  Month 8- Concern about unwanted disclosure of HIV status when attending appointments at the IC?: Missing | 1

59. Secondary Outcome: Number of IC/ASA Staff Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration in Participants With Other Quantitative Questionnaires Prior to Month 1
Description: Since CABENUVA must be administered within a two-week treatment window every month, IC/ASA staff were asked their opinion about the ease or difficulty in appointment re-scheduling and implementation of CABENUVA administration in their work-flow.
Time Frame: Prior to Month 1 (Baseline)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 113
Participants
  How easy or difficult do you think the appointment re-scheduling will be?: Extremely easy | 6
  How easy or difficult do you think the appointment re-scheduling will be?: Very easy | 24
  How easy or difficult do you think the appointment re-scheduling will be?: Somewhat easy | 16
  How easy or difficult do you think the appointment re-scheduling will be?: Neutral | 46
  How easy or difficult do you think the appointment re-scheduling will be?: Somewhat difficult | 15
  How easy or difficult do you think the appointment re-scheduling will be?: Very difficult | 6
  How easy or difficult do you think the appointment re-scheduling will be?: Extremely difficult | 0
  How easy or difficult CABENUVA administration will be to implement in your current work-flow?: Extremely easy | 9
  How easy or difficult CABENUVA administration will be to implement in your current work-flow?: Very easy | 21
  How easy or difficult CABENUVA administration will be to implement in your current work-flow?: Somewhat easy | 21
  How easy or difficult CABENUVA administration will be to implement in your current work-flow?: Neutral | 31
  How easy or difficult CABENUVA administration will be to implement in your current work-flow?: Somewhat difficult | 19
  How easy or difficult CABENUVA administration will be to implement in your current work-flow?: Very difficult | 9
  How easy or difficult CABENUVA administration will be to implement in your current work-flow?: Extremely difficult | 3

60. Secondary Outcome: Number of IC/ASA Staff Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration in Participants With Other Quantitative Questionnaires at Month 3
Description: Since CABENUVA must be administered within a two-week treatment window (+/-)7 days relative to the target treatment date), the IC/ASA staff was asked their opinion about the ease or difficulty in appointment scheduling and re-scheduling and implementation of CABENUVA administration in their workflow.
Time Frame: At Month 3
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 38
Participants
  Ease or difficulty in appointment scheduling for CABENUVA injections-Extremely easy | 2
  Ease or difficulty in appointment scheduling for CABENUVA injections-Very easy | 2
  Ease or difficulty in appointment scheduling for CABENUVA injections-Somewhat easy | 7
  Ease or difficulty in appointment scheduling for CABENUVA injections-Neither easy nor difficult | 6
  Ease or difficulty in appointment scheduling for CABENUVA injections-Somewhat difficult | 2
  Ease or difficulty in appointment scheduling for CABENUVA injections-Very difficult | 0
  Ease or difficulty in appointment scheduling for CABENUVA injections-Extremely difficult | 0
  Ease or difficulty in appointment scheduling for CABENUVA injections-Unsure/not applicable to role | 15
  Ease or difficulty in appointment scheduling for CABENUVA injections- Missing | 4
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Extremely easy: number analyzed (Participants) | 23
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Extremely easy | 1
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Very easy: number analyzed (Participants) | 23
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Very easy | 2
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Somewhat easy: number analyzed (Participants) | 23
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Somewhat easy | 6
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Neither easy nor difficult: number analyzed (Participants) | 23
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Neither easy nor difficult | 5
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Somewhat difficult: number analyzed (Participants) | 23
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Somewhat difficult | 1
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Very difficult: number analyzed (Participants) | 23
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Very difficult | 0
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Extremely difficult: number analyzed (Participants) | 23
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Extremely difficult | 0
  Ease or difficulty in appointment re-scheduling for CABENUVA injections-Unsure/NA to role: number analyzed (Participants) | 23
  Ease or difficulty in appointment re-scheduling for CABENUVA injections-Unsure/NA to role | 4
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Missing: number analyzed (Participants) | 23
  Ease or difficulty in appointment re-scheduling for CABENUVA injections- Missing | 4
  Ease or difficulty in implementation of CABENUVA administration- Extremely easy | 2
  Ease or difficulty in implementation of CABENUVA administration- Very easy | 6
  Ease or difficulty in implementation of CABENUVA administration- Somewhat easy | 3
  Ease or difficulty in implementation of CABENUVA administration- Neither easy nor difficult | 16
  Ease or difficulty in implementation of CABENUVA administration- Somewhat difficult | 4
  Ease or difficulty in implementation of CABENUVA administration- Very difficult | 2
  Ease or difficulty in implementation of CABENUVA administration- Extremely difficult | 1
  Ease or difficulty in implementation of CABENUVA administration- Unsure/not applicable to role | NA — This category is not applicable for this question.
  Ease or difficulty in implementation of CABENUVA administration- Missing | 4

61. Secondary Outcome: Number of IC/ASA Staff Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration in Participants With Other Quantitative Questionnaires at Month 8
Description: as for outcome 60
Time Frame: At Month 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 26
Participants
  How easy or difficult has it been to schedule appointments for CABENUVA injections.: Extremely easy | 2
  How easy or difficult has it been to schedule appointments for CABENUVA injections.: Very easy | 2
  How easy or difficult has it been to schedule appointments for CABENUVA injections.: Somewhat easy | 4
  How easy or difficult has it been to schedule appointments for CABENUVA injections.: Neither easy nor difficult | 1
  How easy or difficult has it been to schedule appointments for CABENUVA injections.: Somewhat difficult | 1
  How easy or difficult has it been to schedule appointments for CABENUVA injections.: Very difficult | 1
  How easy or difficult has it been to schedule appointments for CABENUVA injections.: Extremely difficult | 0
  How easy or difficult has it been to schedule appointments for CABENUVA injections.: Unsure/not applicable to role | 8
  How easy or difficult has it been to schedule appointments for CABENUVA injections.: Missing | 7
  How easy or difficult has it been to reschedule appointments for CABENUVA injections?: number analyzed (Participants) | 18
  How easy or difficult has it been to reschedule appointments for CABENUVA injections?: Extremely easy | 0
  How easy or difficult has it been to reschedule appointments for CABENUVA injections?: Very easy | 6
  How easy or difficult has it been to reschedule appointments for CABENUVA injections?: Somewhat easy | 1
  How easy or difficult has it been to reschedule appointments for CABENUVA injections?: Neither easy nor difficult | 1
  How easy or difficult has it been to reschedule appointments for CABENUVA injections?: Somewhat difficult | 2
  How easy or difficult has it been to reschedule appointments for CABENUVA injections?: Very difficult | 1
  How easy or difficult has it been to reschedule appointments for CABENUVA injections?: Extremely difficult | 0
  How easy or difficult has it been to reschedule appointments for CABENUVA injections?: Unsure/not applicable to role | 1
  How easy or difficult has it been to reschedule appointments for CABENUVA injections?: Missing | 6
  How easy or difficult has CABENUVA administration been to implement in your current work-flow?: Extremely easy | 3
  How easy or difficult has CABENUVA administration been to implement in your current work-flow?: Very easy | 3
  How easy or difficult has CABENUVA administration been to implement in your current work-flow?: Somewhat easy | 2
  How easy or difficult has CABENUVA administration been to implement in your current work-flow?: Neither easy nor difficult | 5
  How easy or difficult has CABENUVA administration been to implement in your current work-flow?: Somewhat difficult | 7
  How easy or difficult has CABENUVA administration been to implement in your current work-flow?: Very difficult | 0
  How easy or difficult has CABENUVA administration been to implement in your current work-flow?: Extremely difficult | 0
  How easy or difficult has CABENUVA administration been to implement in your current work-flow?: Unsure/not applicable to role | NA — This category is not applicable for this question.
  How easy or difficult has CABENUVA administration been to implement in your current work-flow?: Missing | 6

62. Secondary Outcome: Number of HIV Care Providers Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration in Participants With Quantitative Questionnaires at Month 1
Time Frame: At Month 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- HIV Care Provider: Eligible HIV Care Providers completed study assessments at each data collection time point.
Arm/Group | HIV Care Provider
Number analyzed (Participants) | 3
Participants
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Extremely concerned | 1
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Moderately concerned | 1
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Somewhat concerned | 1
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Slightly concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Not at all concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Missing | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Extremely concerned | 1
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Moderately concerned | 1
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Somewhat concerned | 1
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Slightly concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Not at all concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Missing | 0
  Patients not being virologically suppressed due to missed injections: Extremely concerned | 0
  Patients not being virologically suppressed due to missed injections: Moderately concerned | 2
  Patients not being virologically suppressed due to missed injections: Somewhat concerned | 1
  Patients not being virologically suppressed due to missed injections: Slightly concerned | 0
  Patients not being virologically suppressed due to missed injections: Not at all concerned | 0
  Patients not being virologically suppressed due to missed injections: Missing | 0
  Being informed (in a timely manner) of adverse events: Extremely concerned | 0
  Being informed (in a timely manner) of adverse events: Moderately concerned | 2
  Being informed (in a timely manner) of adverse events: Somewhat concerned | 1
  Being informed (in a timely manner) of adverse events: Slightly concerned | 0
  Being informed (in a timely manner) of adverse events: Not at all concerned | 0
  Being informed (in a timely manner) of adverse events: Missing | 0
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Extremely concerned | 0
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Moderately concerned | 2
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Somewhat concerned | 0
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Slightly concerned | 1
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Not at all concerned | 0
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Missing | 0

63. Secondary Outcome: Number of HIV Care Providers Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration in Participants With Quantitative Questionnaires at Month 4
Time Frame: At Month 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Provider
Number analyzed (Participants) | 3
Participants
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Extremely concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Moderately concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Somewhat concerned | 3
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Slightly concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Not at all concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Missing | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Extremely concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Moderately concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Somewhat concerned | 3
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Slightly concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Not at all concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Missing | 0
  Patients not being virologically suppressed due to missed injections: Extremely concerned | 0
  Patients not being virologically suppressed due to missed injections: Moderately concerned | 2
  Patients not being virologically suppressed due to missed injections: Somewhat concerned | 0
  Patients not being virologically suppressed due to missed injections: Slightly concerned | 1
  Patients not being virologically suppressed due to missed injections: Not at all concerned | 0
  Patients not being virologically suppressed due to missed injections: Missing | 0
  Being informed (in a timely manner) of adverse events: Extremely concerned | 0
  Being informed (in a timely manner) of adverse events: Moderately concerned | 1
  Being informed (in a timely manner) of adverse events: Somewhat concerned | 1
  Being informed (in a timely manner) of adverse events: Slightly concerned | 1
  Being informed (in a timely manner) of adverse events: Not at all concerned | 0
  Being informed (in a timely manner) of adverse events: Missing | 0
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Extremely concerned | 1
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Moderately concerned | 0
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Somewhat concerned | 1
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Slightly concerned | 1
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Not at all concerned | 0
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Missing | 0

64. Secondary Outcome: Number of HIV Care Providers Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration in Participants With Quantitative Questionnaires at Month 8
Time Frame: At Month 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Provider
Number analyzed (Participants) | 3
Participants
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Extremely concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Moderately concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Somewhat concerned | 1
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Slightly concerned | 1
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Not at all concerned | 0
  Being informed (in a timely manner) when a patient misses a CABENUVA visit: Missing | 1
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Extremely concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Moderately concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Somewhat concerned | 1
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Slightly concerned | 1
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Not at all concerned | 0
  Infusion Center's (lack of) persistence to follow up with patients on missed appointments: Missing | 1
  Patients not being virologically suppressed due to missed injections: Extremely concerned | 0
  Patients not being virologically suppressed due to missed injections: Moderately concerned | 0
  Patients not being virologically suppressed due to missed injections: Somewhat concerned | 0
  Patients not being virologically suppressed due to missed injections: Slightly concerned | 2
  Patients not being virologically suppressed due to missed injections: Not at all concerned | 0
  Patients not being virologically suppressed due to missed injections: Missing | 1
  Being informed (in a timely manner) of adverse events: Extremely concerned | 0
  Being informed (in a timely manner) of adverse events: Moderately concerned | 0
  Being informed (in a timely manner) of adverse events: Somewhat concerned | 0
  Being informed (in a timely manner) of adverse events: Slightly concerned | 1
  Being informed (in a timely manner) of adverse events: Not at all concerned | 1
  Being informed (in a timely manner) of adverse events: Missing | 1
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Extremely concerned | 0
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Moderately concerned | 0
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Somewhat concerned | 1
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Slightly concerned | 0
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Not at all concerned | 1
  IC's ability to manage other care needs of patients presenting to CABENUVA appointments: Missing | 1

65. Secondary Outcome: Number of Participants Assessed for Facilitators of CABENUVA Administration by Qualitative Interviews at Month 8
Description: Participants were asked about facilitators that made the process of receiving CABENUVA at IC/ASAs easier.
Time Frame: At Month 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 28
Participants
  IC/ASA staff make treatment a positive experience | 8
  Efficiency of treatment | 3
  Clear communication by IC/ASA staff | 5
  Convenience/accessibility of IC/ASA location | 4
  Ease of scheduling appointments and timely reminders | 1
  Not reported | 7

66. Secondary Outcome: Number of IC/ASA Staff Assessed for Barriers/Concerns of CABENUVA Administration in Participants by Qualitative Interviews at Month 8
Description: IC/ASA staff were asked their opinion on the infrastructure impact of administering CABENUVA.
Time Frame: At Month 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 12
Participants
  Facilitates implementation | 12
  Scheduling system work arounds to accommodate visit window | 1
  Modifying visit duration to account for all the pieces of administering CABENUVA | 2
  Shortage of private rooms | 4

67. Secondary Outcome: Number of HIV Care Providers Assessed for Perceptions, Facilitators and Barriers/Concerns of CABENUVA Administration in Participants by Qualitative Interviews at Month 8
Description: HIV care providers were asked about the facilitators and challenges related to referring participants to IC/ASAs.
Time Frame: At Month 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Provider
Number analyzed (Participants) | 3
Participants
  Sending of prescription is not through EMR | 1
  Knowing which IC/ASAs offer CABENUVA | 1
  Multiple labs for participants | 1
  IC/ASA managing insurance | 1
  Participant self-motivation to manage care | 1
  IC/ASA staff support of process | 1

68. Secondary Outcome: Number of Participants Assessed for Preference on the Location to Receive CABENUVA With Other Quantitative Questionnaires at Months 1, 3 and 8
Time Frame: At Month 1, 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 44
Participants
  Month 1- Where would you prefer to receive CABENUVA?: At an infusion center | 28
  Month 1- Where would you prefer to receive CABENUVA?: At home | 8
  Month 1- Where would you prefer to receive CABENUVA?: At my HIV doctor's clinic | 5
  Month 1- Where would you prefer to receive CABENUVA?: At a pharmacy | 2
  Month 1- Where would you prefer to receive CABENUVA?: Other | 0
  Month 1- Where would you prefer to receive CABENUVA?: Missing | 1
  Month 3- Where would you prefer to receive CABENUVA?: number analyzed (Participants) | 41
  Month 3- Where would you prefer to receive CABENUVA?: At an infusion center | 18
  Month 3- Where would you prefer to receive CABENUVA?: At home | 9
  Month 3- Where would you prefer to receive CABENUVA?: At my HIV doctor's clinic | 6
  Month 3- Where would you prefer to receive CABENUVA?: At a pharmacy | 1
  Month 3- Where would you prefer to receive CABENUVA?: Other | 1
  Month 3- Where would you prefer to receive CABENUVA?: Missing | 6
  Month 8- Where would you prefer to receive CABENUVA?: number analyzed (Participants) | 38
  Month 8- Where would you prefer to receive CABENUVA?: At an infusion center | 21
  Month 8- Where would you prefer to receive CABENUVA?: At home | 10
  Month 8- Where would you prefer to receive CABENUVA?: At my HIV doctor's clinic | 3
  Month 8- Where would you prefer to receive CABENUVA?: At a pharmacy | 1
  Month 8- Where would you prefer to receive CABENUVA?: Other | 0
  Month 8- Where would you prefer to receive CABENUVA?: Missing | 3

69. Secondary Outcome: Number of Participants Assessed for Preference on the Location to Receive CABENUVA by Qualitative Interviews at Month 8
Time Frame: At Month 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 33
Participants
  Comfortable with care at IC/ASA | 20
  Home | 5
  Closer proximity to participants | 8

70. Secondary Outcome: Number of Participants Assessed for Advantages of Receiving CABENUVA at IC/ ASA by Other Quantitative Questionnaires at Month 1
Description: In this outcome measure, participants were asked about their views on the IC/ASA administration model (advantages of going to the infusion center to receive CABENUVA).
Time Frame: At Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 44
Participants
  Convenient location of the infusion center | 22
  Ease of parking at the infusion center | 21
  More privacy at the infusion center | 19
  Convenient hours for the infusion center | 17
  Reduced stigma | 13
  I like that people do not know what medication I am there to receive | 12
  Injections are not available at my provider's office | 8
  Other | 2
  No advantages of receiving CABENUVA at the infusion center | 1
  Missing | 1

71. Secondary Outcome: Number of Participants Assessed for Advantages of Receiving CABENUVA at IC/ ASA by Other Quantitative Questionnaires at Months 3 and 8
Description: as for outcome 70
Time Frame: At Months 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 41
Participants
  Month 3- Convenient location of the infusion center | 20
  Month 3- Ease of parking at the infusion center | 19
  Month 3- Ease of scheduling and rescheduling appointments | 17
  Month 3- More privacy at the infusion center | 17
  Month 3- Convenient hours for the infusion center | 13
  Month 3- Reduced stigma | 10
  Month 3- I like that people do not know what medication I am there to receive | 12
  Month 3- Injections are not available at my provider's office | 11
  Month 3- Other | 0
  Month 3- No advantages of receiving CABENUVA at the infusion center | 0
  Month 3- Missing | 5
  Month 8- Convenient location of the infusion center: number analyzed (Participants) | 38
  Month 8- Convenient location of the infusion center | 22
  Month 8- Ease of parking at the infusion center: number analyzed (Participants) | 38
  Month 8- Ease of parking at the infusion center | 24
  Month 8- Ease of scheduling and rescheduling appointments: number analyzed (Participants) | 38
  Month 8- Ease of scheduling and rescheduling appointments | 21
  Month 8- More privacy at the infusion center: number analyzed (Participants) | 38
  Month 8- More privacy at the infusion center | 18
  Month 8- Convenient hours for the infusion center: number analyzed (Participants) | 38
  Month 8- Convenient hours for the infusion center | 13
  Month 8- Reduced stigma: number analyzed (Participants) | 38
  Month 8- Reduced stigma | 16
  Month 8- I like that people do not know what medication I am there to receive: number analyzed (Participants) | 38
  Month 8- I like that people do not know what medication I am there to receive | 18
  Month 8- Injections are not available at my provider's office: number analyzed (Participants) | 38
  Month 8- Injections are not available at my provider's office | 11
  Month 8- Other: number analyzed (Participants) | 38
  Month 8- Other | 3
  Month 8- No advantages of receiving CABENUVA at the infusion center: number analyzed (Participants) | 38
  Month 8- No advantages of receiving CABENUVA at the infusion center | 2
  Month 8- Missing: number analyzed (Participants) | 38
  Month 8- Missing | 1

72. Secondary Outcome: Number of HIV Care Providers Assessed for Advantages of Referring Participants to the IC/ ASA to Receive CABENUVA by Other Quantitative Questionnaires at Month 1, 4 and 8
Description: In this outcome measure, HIV care providers were asked about their views on the IC/ASA administration model (advantages of referring patients to an infusion center for CABENUVA).
Time Frame: At Months 1, 4 and 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 3
Participants
  Month 1- Convenience for the patient | 3
  Month 1- Infusions centers have more clinic space | 1
  Month 1- Infusion centers have more time to add visits to their schedules | 1
  Month 1- Infusion centers have more staff to manage scheduling or rescheduling appointments | 1
  Month 1- Infusion centers have more staff to administer it | 1
  Month 1- Infusion centers have the space to store the medication | 1
  Month 1- Infusion center handles the logistics of administration | 1
  Month 1- Infusion centers manage the insurance verification process | 1
  Month 1- Infusion centers manage acquisition of the medication | 0
  Month 1- Infusion centers manage the insurance reimbursement | 0
  Month 1- Financial considerations for my clinic | 0
  Month 1- Other | 0
  Month 1- Missing | 0
  Month 4- Convenience for the patient | 2
  Month 4- Infusions centers have more clinic space | 1
  Month 4- Infusion centers have more time to add visits to their schedules | 1
  Month 4- Infusion centers have more staff to manage scheduling or rescheduling appointments | 2
  Month 4- Infusion centers have more staff to administer it | 0
  Month 4- Infusion centers have the space to store the medication | 0
  Month 4- Infusion center handles the logistics of administration | 2
  Month 4- Infusion centers manage the insurance verification process | 1
  Month 4- Infusion centers manage acquisition of the medication | 2
  Month 4- Infusion centers manage the insurance reimbursement | 0
  Month 4- Financial considerations for my clinic | 1
  Month 4- Other | 0
  Month 4- Missing | 0
  Month 8- Convenience for the patient | 2
  Month 8- Infusions centers have more clinic space | 1
  Month 8- Infusion centers have more time to add visits to their schedules | 2
  Month 8- Infusion centers have more staff to manage scheduling or rescheduling appointments | 1
  Month 8- Infusion centers have more staff to administer it | 0
  Month 8- Infusion centers have the space to store the medication | 0
  Month 8- Infusion center handles the logistics of administration | 1
  Month 8- Infusion centers manage the insurance verification process | 2
  Month 8- Infusion centers manage acquisition of the medication | 1
  Month 8- Infusion centers manage the insurance reimbursement | 2
  Month 8- Financial considerations for my clinic | 0
  Month 8- Other | 0
  Month 8- Missing | 1

73. Secondary Outcome: Number of Participants Assessed for Advantages of Receiving CABENUVA at IC/ ASA by Qualitative Interviews at Month 8
Time Frame: At Month 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 28
Participants
  Professionalism of staff | 16
  Privacy | 9
  Overall convenience | 14

74. Secondary Outcome: Number of HIV Care Providers Assessed for Advantages of Participants Receiving CABENUVA at IC/ ASA by Qualitative Interviews at Month 8
Time Frame: At Month 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 2
Participants
  Convenience | 2
  Efficiency | 2

75. Secondary Outcome: Number of Participants Assessed for Disadvantages of Receiving CABENUVA at IC/ ASA by Other Quantitative Questionnaires at Month 1
Description: In this outcome measure, participants were asked about their views on the IC/ASA administration model (disadvantages of going to the infusion center to receive CABENUVA).
Time Frame: At Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 44
Participants
  No disadvantages of receiving CABENUVA at the infusion center | 23
  Inconvenient location of the infusion center | 8
  Unfamiliar with routine at the infusion center | 5
  Inconvenient hours for the infusion center | 4
  I don't want other people at the infusion center to know I have HIV | 4
  Decreased contact with my HIV provider | 3
  Too many appointments between the IC and the HIV doctors | 3
  Unfamiliar with the infusion center staff | 2
  Less privacy at the infusion center | 2
  Other | 1
  Difficulty scheduling and rescheduling appointments at the infusion center | 0
  Too many lab draws | 0
  Infusion center doesn't know how to manage the pain or side effects of CABENUVA | 0
  Missing | 1

76. Secondary Outcome: Number of Participants Assessed for Disadvantages of Receiving CABENUVA at IC/ ASA by Other Quantitative Questionnaires at Months 3 and 8
Description: as for outcome 75
Time Frame: At Months 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 41
Participants
  Month 3- No disadvantages of receiving CABENUVA at the infusion center | 16
  Month 3- Inconvenient location of the infusion center | 7
  Month 3- Unfamiliar with routine at the infusion center | 1
  Month 3- Inconvenient hours for the infusion center | 3
  Month 3- I don't want other people at the infusion center to know I have HIV | 6
  Month 3- Decreased contact with my HIV provider | 7
  Month 3- Too many appointments between the IC and the HIV doctors | 2
  Month 3- Unfamiliar with the infusion center staff | 1
  Month 3- Less privacy at the infusion center | 2
  Month 3- Other | 0
  Month 3- Difficulty scheduling and rescheduling appointments at the infusion center | 0
  Month 3- Too many lab draws | 1
  Month 3- Infusion center doesn't know how to manage the pain or side effects of CABENUVA | 1
  Month 3- More stigma at the infusion center | 2
  Month 3- Difficulty of parking at the infusion center | 0
  Month 3- Missing | 7
  Month 8- No disadvantages of receiving CABENUVA at the infusion center: number analyzed (Participants) | 38
  Month 8- No disadvantages of receiving CABENUVA at the infusion center | 17
  Month 8- Inconvenient location of the infusion center: number analyzed (Participants) | 38
  Month 8- Inconvenient location of the infusion center | 8
  Month 8- Unfamiliar with routine at the infusion center: number analyzed (Participants) | 38
  Month 8- Unfamiliar with routine at the infusion center | 0
  Month 8- Inconvenient hours for the infusion center: number analyzed (Participants) | 38
  Month 8- Inconvenient hours for the infusion center | 5
  Month 8- I don't want other people at the infusion center to know I have HIV: number analyzed (Participants) | 38
  Month 8- I don't want other people at the infusion center to know I have HIV | 5
  Month 8- Decreased contact with my HIV provider: number analyzed (Participants) | 38
  Month 8- Decreased contact with my HIV provider | 7
  Month 8- Too many appointments between the IC and the HIV doctors: number analyzed (Participants) | 38
  Month 8- Too many appointments between the IC and the HIV doctors | 1
  Month 8- Unfamiliar with the infusion center staff: number analyzed (Participants) | 38
  Month 8- Unfamiliar with the infusion center staff | 1
  Month 8- Less privacy at the infusion center: number analyzed (Participants) | 38
  Month 8- Less privacy at the infusion center | 3
  Month 8- Other: number analyzed (Participants) | 38
  Month 8- Other | 1
  Month 8- Difficulty scheduling and rescheduling appointments at the infusion center: number analyzed (Participants) | 38
  Month 8- Difficulty scheduling and rescheduling appointments at the infusion center | 0
  Month 8- Too many lab draws: number analyzed (Participants) | 38
  Month 8- Too many lab draws | 1
  Month 8- Infusion center doesn't know how to manage the pain or side effects of CABENUVA: number analyzed (Participants) | 38
  Month 8- Infusion center doesn't know how to manage the pain or side effects of CABENUVA | 0
  Month 8- More stigma at the infusion center: number analyzed (Participants) | 38
  Month 8- More stigma at the infusion center | 1
  Month 8- Difficulty of parking at the infusion center: number analyzed (Participants) | 38
  Month 8- Difficulty of parking at the infusion center | 2
  Month 8- Missing: number analyzed (Participants) | 38
  Month 8- Missing | 1

77. Secondary Outcome: Number of HIV Care Providers Assessed for Disadvantages of Referring Participants to the IC/ ASA to Receive CABENUVA by Other Quantitative Questionnaires at Month 1
Description: In this outcome measure, HIV care providers were asked about their views on the IC/ASA administration model (potential disadvantages of referring patients to an IC for CABENUVA).
Time Frame: At Month 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 3
Participants
  Concern I won't be aware if my patient does not receive CABENUVA on time | 3
  Concern about adverse event management | 2
  Inconvenience for patients to go to two locations (clinic for routine visits and IC for injections) | 2
  Concern about management of injection site reactions | 1
  Concern patient won't want to go to infusion center | 1
  Concern about stigma patient may experience receiving an CABENUVA at infusion center | 1
  Missed opportunity for revenue for my HIV clinic | 1
  Issues with ICs handling logistics associated with insurance verification and approval | 1
  Concern I won't be aware when my patient receives CABENUVA | 0
  Concern about reduced involvement in management of HIV-related care | 0
  Issues with infusion centers handling the logistics associated with insurance reimbursement | 0
  Fear of losing my patient to another provider | 0
  Other | 0
  Missing | 0

78. Secondary Outcome: Number of HIV Care Providers Assessed for Disadvantages of Referring Participants to the IC/ ASA to Receive CABENUVA by Other Quantitative Questionnaires at Months 4 and 8
Description: In this outcome measure, HIV care providers were asked about their views on the IC/ASA administration model (disadvantages of referring patients to an IC for CABENUVA).
Time Frame: At Months 4 and 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 3
Participants
  Month 4- Concern I won't be aware if my patient does not receive CABENUVA on time | 1
  Month 4- Concern about adverse event management | 1
  Month4-Inconvenience for patients to go to 2 locations(clinic for routine visits & IC for injections | 1
  Month 4- Concern about management of injection site reactions | 0
  Month 4- Concern patient won't want to go to infusion center | 0
  Month 4- Concern about stigma patient may experience receiving an CABENUVA at infusion center | 1
  Month 4- Missed opportunity for revenue for my HIV clinic | 1
  Month 4- Issues with ICs handling logistics associated with insurance verification and approval | 0
  Month 4- Concern I won't be aware when my patient receives CABENUVA | 0
  Month 4- Concern about reduced involvement in management of HIV-related care | 2
  Month 4- Issues with infusion centers handling the logistics associated with insurance reimbursement | 0
  Month 4- Fear of losing my patient to another provider | 1
  Month 4- Other | 0
  Month 4- Missing | 0
  Month 8- Concern I won't be aware if my patient does not receive CABENUVA on time | 1
  Month 8- Concern about adverse event management | 0
  Month8-Inconvenience for patients to go to 2 locations(clinic for routine visits & IC for injections | 1
  Month 8- Concern about management of injection site reactions | 0
  Month 8- Concern patient won't want to go to infusion center | 0
  Month 8- Concern about stigma patient may experience receiving an CABENUVA at infusion center | 0
  Month 8- Missed opportunity for revenue for my HIV clinic | 0
  Month 8- Issues with ICs handling logistics associated with insurance verification and approval | 0
  Month 8- Concern I won't be aware when my patient receives CABENUVA | 1
  Month 8- Concern about reduced involvement in management of HIV-related care | 2
  Month 8- Issues with infusion centers handling the logistics associated with insurance reimbursement | 0
  Month 8- Fear of losing my patient to another provider | 0
  Month 8- Other | 0
  Month 8- Missing | 1

79. Secondary Outcome: Number of Participants Assessed for Disadvantages of Receiving CABENUVA at IC/ ASA by Qualitative Interviews at Month 8
Time Frame: At Month 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 28
Participants
  Distance spent traveling to IC/ASA | 17
  Privacy due to traveling outside home for treatment | 3
  Not reported | 8

80. Secondary Outcome: Number of HIV Care Providers Assessed for Disadvantages for Participants Receiving CABENUVA at IC/ ASA by Qualitative Interviews at Month 8
Description: In this outcome measure, HIV care providers were asked about their views on the IC/ASA administration model (disadvantages for participants receiving CABENUVA at IC/ASAs).
Time Frame: At Month 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 2
Participants
  Stigma | 2
  Does not see how it is easier for participants | 1

81. Secondary Outcome: Number of Participants Assessed for Acceptability of the Process of Receiving Injections at ICs/ ASAs by Other Quantitative Questionnaires at Month 1
Time Frame: At Month 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 44
Participants
  How acceptable is it to you to come to the infusion center for CABENUVA?: Very acceptable | 34
  How acceptable is it to you to come to the infusion center for CABENUVA?: Somewhat acceptable | 6
  How acceptable is it to you to come to the infusion center for CABENUVA?: A little acceptable | 0
  How acceptable is it to you to come to the infusion center for CABENUVA?: Neutral | 2
  How acceptable is it to you to come to the infusion center for CABENUVA?: A little unacceptable | 0
  How acceptable is it to you to come to the infusion center for CABENUVA?: Somewhat unacceptable | 1
  How acceptable is it to you to come to the infusion center for CABENUVA?: Very unacceptable | 0
  How acceptable is it to you to come to the infusion center for CABENUVA?: Missing | 1
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Very acceptable | 19
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Somewhat acceptable | 11
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: A little acceptable | 0
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Neutral | 6
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: A little unacceptable | 4
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Somewhat unacceptable | 2
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Very unacceptable | 1
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Missing | 1
  How acceptable is it for you to get labs drawn at the infusion center?: Very acceptable | 32
  How acceptable is it for you to get labs drawn at the infusion center?: Somewhat acceptable | 5
  How acceptable is it for you to get labs drawn at the infusion center?: A little acceptable | 0
  How acceptable is it for you to get labs drawn at the infusion center?: Neutral | 5
  How acceptable is it for you to get labs drawn at the infusion center?: A little unacceptable | 0
  How acceptable is it for you to get labs drawn at the infusion center?: Somewhat unacceptable | 1
  How acceptable is it for you to get labs drawn at the infusion center?: Very unacceptable | 0
  How acceptable is it for you to get labs drawn at the infusion center?: Missing | 1

82. Secondary Outcome: Number of Participants Assessed for Acceptability of the Process of Receiving Injections at ICs/ ASAs by Other Quantitative Questionnaires at Month 3
Time Frame: At Month 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 41
Participants
  How acceptable is it to you to come to the infusion center for CABENUVA?: Very acceptable | 24
  How acceptable is it to you to come to the infusion center for CABENUVA?: Somewhat acceptable | 9
  How acceptable is it to you to come to the infusion center for CABENUVA?: A little acceptable | 1
  How acceptable is it to you to come to the infusion center for CABENUVA?: Neutral | 0
  How acceptable is it to you to come to the infusion center for CABENUVA?: A little unacceptable | 0
  How acceptable is it to you to come to the infusion center for CABENUVA?: Somewhat unacceptable | 1
  How acceptable is it to you to come to the infusion center for CABENUVA?: Very unacceptable | 1
  How acceptable is it to you to come to the infusion center for CABENUVA?: Missing | 5
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Very acceptable | 14
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Somewhat acceptable | 7
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: A little acceptable | 6
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Neutral | 3
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: A little unacceptable | 2
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Somewhat unacceptable | 2
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Very unacceptable | 2
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Missing | 5
  How acceptable is it for you to get labs drawn at the infusion center?: Very acceptable | 27
  How acceptable is it for you to get labs drawn at the infusion center?: Somewhat acceptable | 3
  How acceptable is it for you to get labs drawn at the infusion center?: A little acceptable | 1
  How acceptable is it for you to get labs drawn at the infusion center?: Neutral | 2
  How acceptable is it for you to get labs drawn at the infusion center?: A little unacceptable | 0
  How acceptable is it for you to get labs drawn at the infusion center?: Somewhat unacceptable | 0
  How acceptable is it for you to get labs drawn at the infusion center?: Very unacceptable | 3
  How acceptable is it for you to get labs drawn at the infusion center?: Missing | 5

83. Secondary Outcome: Number of Participants Assessed for Acceptability of the Process of Receiving Injections at ICs/ ASAs by Other Quantitative Questionnaires at Month 8
Time Frame: At Month 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 38
Participants
  How acceptable is it to you to come to the infusion center for CABENUVA?: Very acceptable | 23
  How acceptable is it to you to come to the infusion center for CABENUVA?: Somewhat acceptable | 8
  How acceptable is it to you to come to the infusion center for CABENUVA?: A little acceptable | 1
  How acceptable is it to you to come to the infusion center for CABENUVA?: Neutral | 4
  How acceptable is it to you to come to the infusion center for CABENUVA?: A little unacceptable | 0
  How acceptable is it to you to come to the infusion center for CABENUVA?: Somewhat unacceptable | 1
  How acceptable is it to you to come to the infusion center for CABENUVA?: Very unacceptable | 0
  How acceptable is it to you to come to the infusion center for CABENUVA?: Missing | 1
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Very acceptable | 15
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Somewhat acceptable | 9
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: A little acceptable | 4
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Neutral | 4
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: A little unacceptable | 1
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Somewhat unacceptable | 2
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Very unacceptable | 2
  Acceptability to go to separate places for care (IC for CABENUVA and clinic for HIV appointments)?: Missing | 1
  How acceptable is it for you to get labs drawn at the infusion center?: Very acceptable | 33
  How acceptable is it for you to get labs drawn at the infusion center?: Somewhat acceptable | 1
  How acceptable is it for you to get labs drawn at the infusion center?: A little acceptable | 1
  How acceptable is it for you to get labs drawn at the infusion center?: Neutral | 1
  How acceptable is it for you to get labs drawn at the infusion center?: A little unacceptable | 0
  How acceptable is it for you to get labs drawn at the infusion center?: Somewhat unacceptable | 1
  How acceptable is it for you to get labs drawn at the infusion center?: Very unacceptable | 0
  How acceptable is it for you to get labs drawn at the infusion center?: Missing | 1

84. Secondary Outcome: Number of Participants Assessed for Acceptability of the Process of Receiving Injections at ICs/ ASAs (Time Spent at IC) by Other Quantitative Questionnaires at Months 3 and 8
Time Frame: At Months 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 41
Participants
  Month 3- Not including first visit, how much time have you spent at the IC for your CABENUVA visits?: 1-15 minutes | 1
  Month 3- Not including first visit, how much time have you spent at the IC for your CABENUVA visits?: 16-30 minutes | 17
  Month 3- Not including first visit, how much time have you spent at the IC for your CABENUVA visits?: 31-45 minutes | 15
  Month 3- Not including first visit, how much time have you spent at the IC for your CABENUVA visits?: 46-60 minutes | 2
  Month 3- Not including first visit, how much time have you spent at the IC for your CABENUVA visits?: More than 60 minutes | 1
  Month 3- Not including first visit, how much time have you spent at the IC for your CABENUVA visits?: Missing | 5
  Month 8- Not including first visit, how much time have you spent at the IC for your CABENUVA visits?: number analyzed (Participants) | 38
  Month 8- Not including first visit, how much time have you spent at the IC for your CABENUVA visits?: 1-15 minutes | 4
  Month 8- Not including first visit, how much time have you spent at the IC for your CABENUVA visits?: 16-30 minutes | 10
  Month 8- Not including first visit, how much time have you spent at the IC for your CABENUVA visits?: 31-45 minutes | 12
  Month 8- Not including first visit, how much time have you spent at the IC for your CABENUVA visits?: 46-60 minutes | 10
  Month 8- Not including first visit, how much time have you spent at the IC for your CABENUVA visits?: More than 60 minutes | 1
  Month 8- Not including first visit, how much time have you spent at the IC for your CABENUVA visits?: Missing | 1

85. Secondary Outcome: Number of HIV Care Providers Assessed for Acceptability of the Process of Referring Participants to the IC/ ASA for CABENUVA by Other Quantitative Questionnaires at Months 1, 4 and 8
Description: HIV care providers were asked about the type of patients they found acceptable to refer to an IC to receive CABENUVA.
Time Frame: At Months 1, 4 and 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 3
Participants
  All patients, Month 1 | 1
  All patients, Month 4 | 0
  All patients, Month 8 | 0
  Patients who want to start CABENUVA but prefer not to come to HIV clinic for each injection, Month 1 | 1
  Patients who want to start CABENUVA but prefer not to come to HIV clinic for each injection, Month 4 | 0
  Patients who want to start CABENUVA but prefer not to come to HIV clinic for each injection, Month 8 | 0
  Patients who have had difficulty maintaining their daily oral treatment regimen, Month 1 | 1
  Patients who have had difficulty maintaining their daily oral treatment regimen, Month 4 | 0
  Patients who have had difficulty maintaining their daily oral treatment regimen, Month 8 | 0
  Patients already receiving CABENUVA, Month 1 | 1
  Patients already receiving CABENUVA, Month 4 | 1
  Patients already receiving CABENUVA, Month 8 | 1
  Other, Month 1 | 1
  Other, Month 4 | 1
  Other, Month 8 | 1
  Patients who have concerns about disclosure of their HIV status to others, Month 1 | 0
  Patients who have concerns about disclosure of their HIV status to others, Month 4 | 0
  Patients who have concerns about disclosure of their HIV status to others, Month 8 | 0
  Patients who feel stigmatized by their HIV, Month 1 | 0
  Patients who feel stigmatized by their HIV, Month 4 | 0
  Patients who feel stigmatized by their HIV, Month 8 | 0
  Patients with more chaotic lifestyles (variable work schedules, frequent travel etc), Month 1 | 0
  Patients with more chaotic lifestyles (variable work schedules, frequent travel etc), Month 4 | 0
  Patients with more chaotic lifestyles (variable work schedules, frequent travel etc), Month 8 | 0
  Patients with more structured lifestyles, Month 1 | 0
  Patients with more structured lifestyles, Month 4 | 0
  Patients with more structured lifestyles, Month 8 | 0
  Newly diagnosed (<2 years since diagnosis), Month 1 | 0
  Newly diagnosed (<2 years since diagnosis), Month 4 | 0
  Newly diagnosed (<2 years since diagnosis), Month 8 | 0
  Treatment experienced, Month 1 | 0
  Treatment experienced, Month 4 | 1
  Treatment experienced, Month 8 | 0
  Younger patients (<35 years old), Month 1 | 0
  Younger patients (<35 years old), Month 4 | 0
  Younger patients (<35 years old), Month 8 | 0
  Older patients (>50 years old), Month 1 | 0
  Older patients (>50 years old), Month 4 | 0
  Older patients (>50 years old), Month 8 | 0
  Missing, Month 1 | 0
  Missing, Month 4 | 0
  Missing, Month 8 | 1

86. Secondary Outcome: Number of Participants Assessed for Acceptability of the Process of Receiving Injections at ICs/ ASAs by Qualitative Interviews at Month 8
Description: Participants were asked about their opinion on the acceptability of CABENUVA administration at the IC.
Time Frame: At Month 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 28
Participants
  Good facilities/environment | 8
  Professional and caring staff | 23
  Consistency of providers | 2
  Protects participants' privacy | 14
  Scheduling flexibility | 4
  Appointment reminders | 1
  Quick and easy administration process | 6
  Hassle-free for participants | 1

87. Secondary Outcome: Number of HIV Care Providers Assessed for Acceptability of the Process of Participants Receiving Injections at ICs/ ASAs by Qualitative Interviews at Month 8
Time Frame: At Month 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 2
Participants
  Reinforcing to have it as an option | 1
  Not reported | 1

88. Secondary Outcome: Number of IC/ASA Staff Assessed for Usefulness of the Blueprint Intervention With Other Quantitative Questionnaires Prior to Month 1
Description: The blueprint guides IC/ASA staff on what to do with referrals to receive CABENUVA at the IC/ASA.
Time Frame: Prior to Month 1 (Baseline)
Population: Analysis was planned to be performed on the IC/ASA staff which includes any IC/ASA staff who completed any portion of any questionnaire at the specified timepoint. Prior to Month 1 there were no referrals given; hence the blueprint was not used and therefore it was not assessed.
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 0

89. Secondary Outcome: Number of IC/ASA Staff Assessed for Usefulness of the Blueprint Intervention With Other Quantitative Questionnaires at Month 3 and 8
Description: The blueprint guides IC/ASA staff on what to do with referrals to receive CABENUVA at the IC/ASA.
Time Frame: At Months 3 and 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 20
Participants
  At month 3 - How useful is the blueprint?: Extremely useful | 2
  At month 3 - How useful is the blueprint?: Very useful | 6
  At month 3 - How useful is the blueprint?: Somewhat useful | 7
  At month 3 - How useful is the blueprint?: Neutral | 4
  At month 3 - How useful is the blueprint?: Not very useful | 0
  At month 3 - How useful is the blueprint?: Not useful at all | 1
  At month 8 - How useful is the blueprint?: number analyzed (Participants) | 15
  At month 8 - How useful is the blueprint?: Extremely useful | 2
  At month 8 - How useful is the blueprint?: Very useful | 3
  At month 8 - How useful is the blueprint?: Somewhat useful | 5
  At month 8 - How useful is the blueprint?: Neutral | 2
  At month 8 - How useful is the blueprint?: Not very useful | 2
  At month 8 - How useful is the blueprint?: Not useful at all | 1

90. Secondary Outcome: Number of HIV Care Providers Assessed for Usefulness of Plan of Treatment (POT) by Other Quantitative Questionnaires at Months 4 and 8
Time Frame: At Months 4 and 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 2
Participants
  Month 4- Information in the POT is comprehensive enough for IC to administer CABENUVA to patients: Strongly Agree | 0
  Month 4- Information in the POT is comprehensive enough for IC to administer CABENUVA to patients: Agree | 2
  Month 4- Information in the POT is comprehensive enough for IC to administer CABENUVA to patients: Occasionally | 0
  Month 4- Information in the POT is comprehensive enough for IC to administer CABENUVA to patients: Neither agree nor disagree | 0
  Month 4- Information in the POT is comprehensive enough for IC to administer CABENUVA to patients: Disagree | 0
  Month 4- Information in the POT is comprehensive enough for IC to administer CABENUVA to patients: Strongly disagree | 0
  Month 4- The POT has all information it should have for the infusion center to administer CABENUVA: Strongly Agree | 1
  Month 4- The POT has all information it should have for the infusion center to administer CABENUVA: Agree | 1
  Month 4- The POT has all information it should have for the infusion center to administer CABENUVA: Occasionally | 0
  Month 4- The POT has all information it should have for the infusion center to administer CABENUVA: Neither agree nor disagree | 0
  Month 4- The POT has all information it should have for the infusion center to administer CABENUVA: Disagree | 0
  Month 4- The POT has all information it should have for the infusion center to administer CABENUVA: Strongly disagree | 0
  Month 8- Information in the POT is comprehensive enough for IC to administer CABENUVA to patients: number analyzed (Participants) | 1
  Month 8- Information in the POT is comprehensive enough for IC to administer CABENUVA to patients: Strongly Agree | 1
  Month 8- Information in the POT is comprehensive enough for IC to administer CABENUVA to patients: Agree | 0
  Month 8- Information in the POT is comprehensive enough for IC to administer CABENUVA to patients: Occasionally | 0
  Month 8- Information in the POT is comprehensive enough for IC to administer CABENUVA to patients: Neither agree nor disagree | 0
  Month 8- Information in the POT is comprehensive enough for IC to administer CABENUVA to patients: Disagree | 0
  Month 8- Information in the POT is comprehensive enough for IC to administer CABENUVA to patients: Strongly disagree | 0
  Month 8- The POT has all information it should have for the infusion center to administer CABENUVA: number analyzed (Participants) | 1
  Month 8- The POT has all information it should have for the infusion center to administer CABENUVA: Strongly Agree | 1
  Month 8- The POT has all information it should have for the infusion center to administer CABENUVA: Agree | 0
  Month 8- The POT has all information it should have for the infusion center to administer CABENUVA: Occasionally | 0
  Month 8- The POT has all information it should have for the infusion center to administer CABENUVA: Neither agree nor disagree | 0
  Month 8- The POT has all information it should have for the infusion center to administer CABENUVA: Disagree | 0
  Month 8- The POT has all information it should have for the infusion center to administer CABENUVA: Strongly disagree | 0

91. Secondary Outcome: Number of IC/ASA Staff Assessed for Usefulness of the Blueprint Intervention and POT Assessed by Qualitative Interviews at Month 8
Time Frame: Month 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 12
Participants
  Usefulness of the blueprint - Usage | 2
  Usefulness of the blueprint - Familiarity | 3
  Usefulness of the blueprint- Not reported | 7
  Usefulness of POT - Usage | 1
  Usefulness of POT- Not reported | 11

92. Secondary Outcome: Number of HIV Care Providers Assessed for Usefulness of the Blueprint Intervention and POT by Qualitative Interviews at Month 8
Description: The blueprint guides HIV care providers on what to do with referrals to receive CABENUVA at the IC/ASA.
Time Frame: Month 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 2
Participants
  Usefulness of POT: Sufficient in providing information to the IC/ASA | 1
  Usefulness of POT: Not reported | 1
  Usefulness of blueprint: Sufficient in providing information to the IC/ASA | 0
  Usefulness of blueprint: Not reported | 2

93. Secondary Outcome: Number of IC/ASA Staff Assessed for Overall Opinion of Administering the Injection at an IC/ ASA by Other Quantitative Questionnaires Prior to Month 1 and at Months 3 and 8
Time Frame: Prior to Month 1 (Baseline) and Months 3 and 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 113
Participants
  Baseline- Overall opinion about administering CABENUVA for participants at your infusion center?: Extremely positive | 14
  Baseline- Overall opinion about administering CABENUVA for participants at your infusion center?: Very positive | 21
  Baseline- Overall opinion about administering CABENUVA for participants at your infusion center?: Somewhat positive | 21
  Baseline- Overall opinion about administering CABENUVA for participants at your infusion center?: Neutral | 37
  Baseline- Overall opinion about administering CABENUVA for participants at your infusion center?: Somewhat negative | 15
  Baseline- Overall opinion about administering CABENUVA for participants at your infusion center?: Very negative | 3
  Baseline- Overall opinion about administering CABENUVA for participants at your infusion center?: Extremely negative | 1
  Baseline- Overall opinion about administering CABENUVA for participants at your infusion center?: Missing | 1
  Month 3- Overall opinion about administering CABENUVA for participants at your infusion center?: number analyzed (Participants) | 38
  Month 3- Overall opinion about administering CABENUVA for participants at your infusion center?: Extremely positive | 3
  Month 3- Overall opinion about administering CABENUVA for participants at your infusion center?: Very positive | 6
  Month 3- Overall opinion about administering CABENUVA for participants at your infusion center?: Somewhat positive | 3
  Month 3- Overall opinion about administering CABENUVA for participants at your infusion center?: Neutral | 17
  Month 3- Overall opinion about administering CABENUVA for participants at your infusion center?: Somewhat negative | 5
  Month 3- Overall opinion about administering CABENUVA for participants at your infusion center?: Very negative | 0
  Month 3- Overall opinion about administering CABENUVA for participants at your infusion center?: Extremely negative | 0
  Month 3- Overall opinion about administering CABENUVA for participants at your infusion center?: Missing | 4
  Month 8- Overall opinion about administering CABENUVA for participants at your infusion center?: number analyzed (Participants) | 26
  Month 8- Overall opinion about administering CABENUVA for participants at your infusion center?: Extremely positive | 4
  Month 8- Overall opinion about administering CABENUVA for participants at your infusion center?: Very positive | 3
  Month 8- Overall opinion about administering CABENUVA for participants at your infusion center?: Somewhat positive | 5
  Month 8- Overall opinion about administering CABENUVA for participants at your infusion center?: Neutral | 7
  Month 8- Overall opinion about administering CABENUVA for participants at your infusion center?: Somewhat negative | 0
  Month 8- Overall opinion about administering CABENUVA for participants at your infusion center?: Very negative | 0
  Month 8- Overall opinion about administering CABENUVA for participants at your infusion center?: Extremely negative | 0
  Month 8- Overall opinion about administering CABENUVA for participants at your infusion center?: Missing | 7

94. Secondary Outcome: Number of Participants Assessed for Overall Opinion of Receiving the Injection at an IC/ ASA by Other Quantitative Questionnaires at Months 1, 3 and 8
Time Frame: At Months 1, 3 and 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 44
Participants
  At month 1 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Very positive | 35
  At month 1 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Somewhat positive | 5
  At month 1 - What is your overall opinion about going to an infusion center to receive CABENUVA?: A little positive | 1
  At month 1 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Neutral | 1
  At month 1 - What is your overall opinion about going to an infusion center to receive CABENUVA?: A little negative | 1
  At month 1 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Somewhat negative | 0
  At month 1 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Very negative | 0
  At month 1 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Missing | 1
  At month 3 - What is your overall opinion about going to an infusion center to receive CABENUVA?: number analyzed (Participants) | 41
  At month 3 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Very positive | 28
  At month 3 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Somewhat positive | 7
  At month 3 - What is your overall opinion about going to an infusion center to receive CABENUVA?: A little positive | 1
  At month 3 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Neutral | 0
  At month 3 - What is your overall opinion about going to an infusion center to receive CABENUVA?: A little negative | 0
  At month 3 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Somewhat negative | 0
  At month 3 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Very negative | 0
  At month 3 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Missing | 5
  At month 8 - What is your overall opinion about going to an infusion center to receive CABENUVA?: number analyzed (Participants) | 38
  At month 8 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Very positive | 27
  At month 8 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Somewhat positive | 9
  At month 8 - What is your overall opinion about going to an infusion center to receive CABENUVA?: A little positive | 0
  At month 8 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Neutral | 0
  At month 8 - What is your overall opinion about going to an infusion center to receive CABENUVA?: A little negative | 1
  At month 8 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Somewhat negative | 0
  At month 8 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Very negative | 0
  At month 8 - What is your overall opinion about going to an infusion center to receive CABENUVA?: Missing | 1

95. Secondary Outcome: Number of HIV Care Providers Assessed for Overall Opinion of Referring the Participant to an IC/ ASA by Other Quantitative Questionnaires at Month 1
Time Frame: At Month 1
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 3
Participants
  Always | 0
  Often | 1
  Occasionally | 1
  Rarely | 1
  Never | 0
  Missing | 0

96. Secondary Outcome: Number of HIV Care Providers Assessed for Overall Opinion of Referring the Participant to an IC/ ASA by Other Quantitative Questionnaires at Month 4
Time Frame: At Month 4
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 3
Participants
  Very acceptable | 2
  Somewhat acceptable | 1
  A little acceptable | 0
  Neutral | 0
  A little unacceptable | 0
  Somewhat unacceptable | 0
  Very unacceptable | 0
  I have not interacted with the infusion center yet. | 0
  Missing | 0

97. Secondary Outcome: Number of HIV Care Providers Assessed for Overall Opinion of Referring the Participant to an IC/ ASA by Other Quantitative Questionnaires at Month 8
Time Frame: At Month 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 3
Participants
  Extremely satisfied | 0
  Very satisfied | 2
  Somewhat satisfied | 0
  Neutral | 0
  Somewhat dissatisfied | 0
  Very dissatisfied | 0
  Extremely dissatisfied | 0
  I was not involved in this process | 0
  Missing | 1

98. Secondary Outcome: Number of HIV Care Providers Assessed for Overall Opinion of Continuing to Refer Participants to an IC/ ASA by Other Quantitative Questionnaires at Month 8
Time Frame: At Month 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 3
Participants
  Extremely likely | 0
  Very likely | 1
  Somewhat likely | 1
  Neutral | 0
  Somewhat unlikely | 0
  Very unlikely | 0
  Extremely unlikely | 0
  I was not involved in this process | 0
  Missing | 1

99. Secondary Outcome: Number of Participants Assessed for Overall Opinion of Receiving the Injection at an IC/ ASA by Qualitative Interview at Month 8
Description: Participants were asked about their overall favorable and non-favorable opinion of receiving CABENUVA at the IC/ASA.
Time Frame: At Month 8
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 28
Participants
  Effectiveness of treatment | 5
  Convenience of treatment | 11
  No daily reminder of diagnosis | 5
  Treatment cadence | 13
  Not needing to worry about forgetting to take the pill | 5
  Reduced worry about unwanted disclosure of HIV | 4
  Reduces pill burden | 6
  No more pill side effects | 2

100. Secondary Outcome: Number of HIV Care Providers Assessed for Overall Opinion of Referring Patients to an IC/ ASA by Qualitative Interview at Month 8
Description: HIV care providers were asked about their overall favoring and non-favoring opinions on referring participants to IC/ASA for CABENUVA administration.
Time Frame: At Month 8
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV Care Providers
Number analyzed (Participants) | 2
Participants
  Alternative treatment option for participants | 1
  Advantages of CABENUVA over daily pill regimen | 2
  Lack of effectiveness | 1
  Painful for participants | 1
  Injection location on participant | 1

101. Secondary Outcome: Number of IC/ASA Staff Assessed for Overall Opinion of Administering the Injection at an IC/ ASA by Qualitative Interview at Month 8
Description: IC/ASA staff was asked about their overall opinion on the participants referral process.
Time Frame: At Month 8
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | IC/ASA Staff
Number analyzed (Participants) | 12
Participants
  Clinical staff not involved | 12
  Field questions from participants regarding referring friends | 1

102. Secondary Outcome: Number of Injections Occurring Within Target Window From Target Date
Description: This outcome measure evaluates the fidelity to treatment and dosing window. Fidelity to treatment and dosing window was defined based on a ±7-day window from target treatment date based on the calendar date of baseline injection.
Time Frame: Up to and including Month 8
Population: as for outcome 1
Measure: Count of Units; unit: Injections
Units Other Than Participants: Injections
Arm/Group | Participants Receiving CABENUVA
Number analyzed (Participants) | 44
Number analyzed (Injections) | 195
Injections
  <-14 days | 0
  -14 to -8 days | 3
  -7 to -4 days | 37
  -3 to -2 days | 27
  -1 day | 9
  0 day | 36
  1 day | 16
  2 to 3 days | 24
  4 to 7 days | 38
  8 to 14 days | 3
  >14 days | 1
  Missed injection | 1

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and other adverse events (AEs) were reported from Month 1 (signing of informed consent) to Month 8 (study completion).
Description: SAEs, solicited AEs and unsolicited AEs were reported for the Safety set.
Arm/Group | Participants Receiving CABENUVA
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 13/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Receiving CABENUVA (N=44)
Injection site discomfort (General disorders) | 6 (8)
Injection site pain (General disorders) | 6 (7)
Fatigue (General disorders) | 1 (2)
Injection site nodule (General disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-03-29): https://cdn.clinicaltrials.gov/large-docs/45/NCT04982445/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT04982445/SAP_001.pdf